Protocol: MTI-106

- **Protocol number:** MTI-106.
- **Document title:** A randomized, double-blind, placebo-controlled study of the efficacy, safety, and tolerability of serlopitant for the treatment of pruritus in adults with prurigo nodularis.
- Version number: SAP Version 4.
- Date of the document: 16 December 2019.
- NCT number: NCT03677401

# STATISTICAL ANALYSIS PLAN

Protocol Number: MTI-106

Study Title: A RANDOMIZED, DOUBLE-BLIND, PLACEBO-

CONTROLLED STUDY OF THE EFFICACY,

SAFETY, AND TOLERABILITY OF

SERLOPITANT FOR THE TREATMENT OF PRURITUS IN ADULTS WITH PRURIGO

**NODULARIS** 

Development Phase of Study: Phase 3

Sponsor: Menlo Therapeutics Inc.

200 Cardinal Way, 2<sup>nd</sup> Floor Redwood City, CA 94063

USA

Sponsor Contact: PPD

Statistical Analysis Plan based on

Protocol Version:

Version 4.0, 16 December 2019

Statistical Analysis Plan Date: 16 December 2019

Statistical Analysis Plan Version: Version 4

Confidentiality Statement:

This document is a confidential communication of Menlo Therapeutics Inc. As such, the recipients agree not to disclose or reproduce, without prior written approval, this document and any attachments, except to appropriate Institutional Review Boards, Ethics Committees, representatives of the US Food and Drug Administration, other regulatory agencies or as otherwise required by applicable laws or regulations.

| Authored by: | |
|--------------|-----|
| | PPD |
| Reviewed by: | PPD |
| | FFD |
| | nnn |
| | PPD |

Revisions to the Statistical Analysis Plan described herein must be approved through a formal written amendment with the exception of minor editorial changes to tables, figures, or listing shells, and any necessary textual clarifications for programmers that do not affect the stated analysis variables, study endpoints, or statistical methods.

# TABLE OF CONTENTS

| 1. | LIS | T OF A | ABBREVIATIONS AND DEFINITIONS OF TERMS | 6 |
|---|---|---|---|---|
| 2. | INT | RODU | ICTION | 7 |
| 3. | STU | J <b>DY O</b> l | BJECTIVES | 7 |
| 4. | STUDY DESIGN | | | 7 |
| | 4.1 | Overa | ll Study Design | 7 |
| | | 4.1.1 | Schedule of Visits and Assessments | 8 |
| | | 4.1.2 | Method of Assigning Subjects to Treatment Groups | 8 |
| | | 4.1.3 | Blinding | 8 |
| 5. | EFI | FICAC | Y AND SAFETY ENDPOINTS | 8 |
| | 5.1 | Effica | cy Endpoints | 8 |
| | | 5.1.1 | Primary Efficacy Endpoint | 8 |
| | | 5.1.2 | Key Secondary Efficacy Endpoints | 8 |
| | | 5.1.3 | Additional Secondary Efficacy Endpoints | |
| | 5.2 | Safety | Endpoints | 9 |
| 6. | STA | ATISTI | CAL AND ANALYTICAL PLANS | 9 |
| | 6.1 | Genera | al Methodology | 9 |
| | | 6.1.1 | Statistical Analysis | 10 |
| | | 6.1.2 | Baseline Definition | 10 |
| | | 6.1.3 | Visit Windowing | 10 |
| | | 6.1.4 | Adjustments for Covariates | 11 |
| | | 6.1.5 | Handling of Dropouts or Missing Data | 11 |
| | | 6.1.6 | Interim Analyses and Data Monitoring | 13 |
| | | 6.1.7 | Multicenter Studies | 13 |
| | | 6.1.8 | Multiple Comparisons/Multiplicity | 13 |
| | | 6.1.9 | Examination of Subgroups | 13 |
| | 6.2 | Dispos | sition of Subjects | 13 |
| | 6.3 | Protoc | col Deviations | 13 |
| | 6.4 | Data S | Sets Analyzed | 13 |
| | | 6.4.1 | Intent-to-Treat (ITT) Population | 14 |
| | | 6.4.2 | Safety Population | 14 |
| | | 6.4.3 | Per Protocol Population | 14 |
| | 6.5 | Demo | graphic and Other Baseline Characteristics | 15 |
| | 6.6 | Prior a | and Concomitant Medications | 15 |
| | 6.7 | Analys | sis of Efficacy | 15 |

| | | 6.7.1 | Primary 1 | Efficacy Analysis | 15 |
|---|---|---|---|---|---|
| | | 6.7.2 | Key Seco | ondary Efficacy Analysis | 16 |
| | | 6.7.3 | Addition | al Secondary Efficacy Analysis | 16 |
| | 6.8 | Sensiti | vity Analy | sis | 16 |
| | | 6.8.1 | Last Obs | ervation Carried Forward | 16 |
| | | 6.8.2 | Repeated | Measures Analysis | 16 |
| | | 6.8.3 | Tipping I | Point Analysis | 17 |
| | 6.9 | Safety | Evaluation | 1 | 17 |
| | | 6.9.1 | Extent of | Exposure | 17 |
| | | 6.9.2 | Adverse | Events | 18 |
| | | 6.9.3 | Clinical 1 | Laboratory Evaluation | 18 |
| | | 6.9.4 | Other Ob | servations Related to Safety | 18 |
| | | | 6.9.4.1 | ECG Measurements | 18 |
| | | | 6.9.4.2 | Vital Signs | 19 |
| | | | 6.9.4.3 | Physical Exams | 19 |
| | | | 6.9.4.4 | Menstrual Diaries | 19 |
| | | | 6.9.4.5 | Hospital Anxiety and Depression Scale (HADS) | 19 |
| | | | 6.9.4.6 | Epworth Sleepiness Scale (ESS) | 19 |
| | 6.10 | ) Pharm | acokinetic | Analysis | 19 |
| 7. | DE | ΓERMI | NATION | OF SAMPLE SIZE | 19 |
| 8. | CH. | ANGES | S IN THE | PLANNED ANALYSES | 20 |
| 9. | REI | FEREN | <b>CES</b> | | 20 |
| 10. | IND | EX OF | PLANNE | D END-OF-TEXT TABLES AND FIGURES | 21 |
| 11. | IND | EX OF | ' PLANNE | D LISTINGS | 116 |

# **Revision History:**

| Version | Date | Summary of Changes | Author |
|---|---|---|---|
| Version 1 | 13 November 2018 | Original document | Brian Armstrong |
| Version 2 | 03 April 2019 | Updated title page to reflect current version of protocol. Updated SAP version and date. | Brian Armstrong |
| | | Sections 5.1.2 and 6.1.8 (previously 6.1.7), 6.7.2, 6.8.2 updated to remove Day 7 and Day 3 key secondary endpoints. | |
| | | Section 6.1 updated, Section 6.1.6 added to reflect potential interim analysis. | |
| | | Section 6.1.3, 6.1.5, 6.7 updated to include Week 1 for WI-NRS data. | |
| | | Sections $6.1.6 - 6.1.9$ renumbered to allow for additional section added as $6.1.6$ . | |
| | | Section 7 updated sample size per Phase 2 information. | |
| Version 3 | 30 August 2019 | Updated SAP version and date. | Brian Armstrong |
| | | Editorial and grammatical updates including abbreviations and references. | |
| | | DLQI Question 1 included as Additional Seconary Endpoint; modified changes to planned analysis section. | |
| | | Clarified visit nomenclature for follow-up period. | |
| | | Modified language to indicate no interim analysis will be performed. | |
| | | Added subgroup summaries of primary efficacy endpoint. | |
| | | Added table, figure and listing shells. | |

| Version 4 | 16 December 2019 | Updated SAP version and date. | Brian Armstrong |
|---|---|---|---|
| | | Modified WI-NRS Weekly average computation to require a minimum of 4 values to compute average. | |
| | | DLQI moved from Key Secondary Endpoint to Additional Secondary Endpoint; removed multiple imputation of DLQI. | |
| | | WI-NRS 4-point responder at Week 2 added as Key Secondary Endpoint. | |
| | | Updated changes to planned analysis section to reflect no changes, as protocol was amended. | |
| | | Updated table, figure and listing shells. | |

#### 1. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AE(s) Adverse event(s)
ANCOVA Analysis of covariance
CMH Cochran-Mantel-Haenszel

DLQI Dermatology Life Quality Index

ECG Electrocardiogram eDiary Electronic diary

ESS Epworth Sleepiness Scale

HADS Hospital Anxiety and Depression Scale

IGA PN-A Investigator's Global Assessment of Prurigo Nodularis Activity
IGA PN-S Investigator's Global Assessment of Prurigo Nodularis Stage

ITT Intent-to-treat

LOCF Last observation carried forward

MedDRA Medical Dictionary for Regulatory Activities

MCMC Markov Chain Monte Carlo

PN Prurigo Nodularis

PP Per Protocol

SAE(s) Serious adverse event(s)

SAS® Statistical Analysis System (SAS® Institute Inc., Cary, NC)

TEAE(s) Treatment-emergent adverse event(s)

WHO-DDE World Health Organization Drug Dictionary Enhanced

WI-NRS Worst-Itch Numeric Rating Scale

#### 2. INTRODUCTION

Prurigo nodularis (PN) is a distinctive and easily diagnosable chronic skin condition characterized by the presence of multiple highly pruritic and often symmetrically distributed nodules and papules on the skin (Jorizzo 1981). The nodules and papules in PN can range in size from approximately 0.5 to 3.0 cm and often appear hyperkeratotic, sometimes crateriform, in appearance. Plaques are occasionally present, and the lesions of PN frequently exhibit other features secondary to prolonged and severe scratching behavior, such as post-inflammatory hyperpigmentation, erosion, ulceration, crusting, and bleeding (Zeidler 2016).

Menlo Therapeutics Inc. is pursuing the development of serlopitant for treatment of itch. The MTI-106 study described herein is a double-blind, randomized, placebo-controlled study to assess the efficacy, safety, and tolerability of serlopitant for the treatment of pruritus in adults with PN.

#### 3. STUDY OBJECTIVES

The efficacy objective of this study is to assess the efficacy of serlopitant for the treatment of pruritus in adults with PN.

The safety objective of this study is to assess the safety and tolerability of repeated oral doses of serlopitant in adults with PN.

#### 4. STUDY DESIGN

#### 4.1 Overall Study Design

This is a double-blind, randomized, placebo-controlled study to assess the efficacy, safety, and tolerability of serlopitant for the treatment of pruritus in adults with PN. The study will be conducted at approximately 50 study sites. Subjects who meet the study entry criteria will be randomized in a 1:1 ratio to receive daily oral doses of serlopitant 5 mg or placebo for 10 weeks. After completion of the treatment period or early discontinuation of study drug treatment, all subjects will enter a 3 or 5-week follow-up period. The required follow-up period is defined as a minimum of 3 weeks for those subjects who will enroll in the one-year open-label safety study (MTI-107) on the date of the follow-up visit, and as 5 weeks for those subjects who will not be enrolled in the one-year open-label safety study of serlopitant. Should a subject present for the follow-up visit prior to 5 weeks after the last dose of study drug and be excluded from participation in the one-year study for any reason, the subject will be required to return at 5 weeks after the last dose of study drug for a complete follow-up visit.

This study will consist of three periods, for a total study period of 15-19 weeks:

• Screening period: 2-4 weeks

• Treatment period: 10 weeks

• Follow-up period: 3 or 5 weeks

#### 4.1.1 Schedule of Visits and Assessments

The schedule of assessments can be found in Section 6.5 and Appendix A of the Protocol.

### 4.1.2 Method of Assigning Subjects to Treatment Groups

Eligible subjects will be randomized to receive serlopitant 5 mg or placebo in a 1:1 ratio. Stratified permuted block randomization will be used. Randomization will be stratified by the subject's reported Worst-Itch Numeric Rating Scale (WI-NRS) score for the 1-week period prior to the Baseline visit (6.5 to < 9, 9 to 10).

An interactive web response system will be used to perform the randomization.

### 4.1.3 Blinding

This study will be conducted as a double-blind study with the treatment assignment concealed from the subjects, the investigators and their staff, the Sponsor, and any designees of the Sponsor as required. The placebo will be formulated to be indistinguishable from the active study product(s). Study materials will be packaged and issued in a manner designed to maintain the blind for subjects and all study personnel involved in the direction and execution of study procedures, study assessments, and collection of data. The randomization code for each subject will be available to the sites for use only in an emergency situation. For details of the procedure for unblinding of individual subjects in cases of emergency see Section 7.6 of the Protocol and the Blinding Plan.

#### 5. EFFICACY AND SAFETY ENDPOINTS

#### 5.1 Efficacy Endpoints

### 5.1.1 Primary Efficacy Endpoint

The primary efficacy endpoint is the WI-NRS 4-point responder rate at Week 10.

#### **5.1.2** Key Secondary Efficacy Endpoints

The key secondary efficacy endpoints are as follows:

• The WI-NRS 4-point responder rate at Week 4

• The WI-NRS 4-point responder rate at Week 2

# 5.1.3 Additional Secondary Efficacy Endpoints

Additional secondary efficacy endpoints include the following:

- Change from baseline in WI-NRS to Weeks 2, 4, 6 and 8
- WI-NRS 3-point responder rate at Weeks 2, 4 and 10
- Change from baseline in Investigator's Global Assessment of PN Activity (IGA PN-A) to Weeks 2, 4, 10
- Change from baseline in Investigator's Global Assessment of PN Stage (IGA PN-S) to Weeks 2, 4, 10
- Change from baseline in Dermatology Life Quality Index (DLQI) to Week 10
- Change from baseline in DLQI Question 1 to Week 10

# 5.2 Safety Endpoints

Safety endpoints include the following:

- Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs)
- Changes from baseline in clinical laboratory parameters following study drug exposure
- Changes from baseline in vital sign and electrocardiogram (ECG) parameters following study drug exposure
- Change from baseline in the Hospital Anxiety and Depression Scale (HADS)
- Change from baseline in the Epworth Sleepiness Scale (ESS)

#### 6. STATISTICAL AND ANALYTICAL PLANS

#### 6.1 General Methodology

All statistical processing will be performed using SAS® Version 9.3 or later, unless otherwise stated. Endpoints will be summarized with descriptive statistics by treatment group and visit. For continuous variables, the following information will be presented: n (number of subjects), mean, standard deviation (SD), median, minimum and maximum. For categorical variables, counts and percentages will be used.

Reported adverse events (AEs), medical history, and prior and concomitant procedures and therapies will be classified on the basis of Medical Dictionary for Regulatory Activities

Statistical Analysis Plan for Menlo Therapeutics Inc.
Protocol Number: MTI-106

16 December 2019

(MedDRA) terminology. Concomitant medications will be classified on the basis of World Health Organization Drug Dictionary Enhanced (WHO-DDE) terminology.

#### 6.1.1 Statistical Analysis

All summary tables and data listings will be prepared by QST Consultations, Ltd., utilizing SAS® Version 9.3 or later software. All relevant data collected within the CRF will be included in data listings.

The standard operating procedures of QST Consultations, Ltd. will be followed in the creation and quality control of all data displays.

#### **6.1.2** Baseline Definition

Baseline, for measures other than those collected daily, will be the last recorded value prior to the start of treatment. For daily WI-NRS data captured via electronic diary (eDiary), baseline will be the average result measured over the 7 days prior to treatment.

### 6.1.3 Visit Windowing

Data will be summarized based on nominal visit indications. Data collected during post-treatment follow-up will be summarized as

| Protocol<br>Version(s) | Nominal Visit | Analysis Visit |
|------------------------|------------------|------------------|
| V2.0; V2.1 | 3-Week Follow-up | 3-Week Follow-up |
| V2.0; V2.1 | 5-Week Follow-up | 5-Week Follow-up |

In addition, a "Latest Follow-up" visit will be summarized, which will include the latest available follow-up information for each subject from the 3-, 5- Week Follow-up visits.

Information collected at early treatment discontinuation visits will be mapped to the most appropriate visit based on the midpoints between scheduled visits.



For example, if a subject terminates use of study drug on or after Day 22 but before Day 36, data collected at the early end of treatment visit will be mapped to the Week 4 evaluation for summaries. If the subject has Week 4 values present, the data collected at the early end of

treatment visit will not replace the data collected at Week 4. For the sensitivity efficacy analyses, last observation carried forward (LOCF) will be applied subsequent to mapping the information to the appropriate visit.

Additionally, WI-NRS will be summarized at Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 and 3- and 5- Week Follow-up by averaging the daily results for the 7 days prior to each week. The weekly average values will be calculated if a subject has at least four responses during the 7 day range, as defined below:

| Week/Visit | Study Day Range |
|------------------|----------------------------------------------|
| Week 1 | 2-7 (as Day 1 may be pre or post first dose) |
| Week 2 | 8-14 |
| Week 3 | 15-21 |
| Week 4 | 22-28 |
| Week 5 | 29-35 |
| Week 6 | 36-42 |
| Week 7 | 43-49 |
| Week 8 | 50-56 |
| Week 9 | 57-63 |
| Week 10 | 64-70 |
| 3-Week Follow-up | Post-treatment days 15-21 |
| 5-Week Follow-up | Post-treatment days 29-35 |

# **6.1.4** Adjustments for Covariates

Analysis of covariance will include baseline value as a covariate.

#### 6.1.5 Handling of Dropouts or Missing Data

Should a determination of treatment period (on treatment, pre-treatment, post-treatment) be required for AEs or concomitant medication but the corresponding date is missing, or is a partial date, the event/medication will be considered on treatment unless the portions of the date that are available indicate this is not possible.

The primary method of handling missing efficacy data will be Markov Chain Monte Carlo (MCMC) multiple imputation. Imputation will be conducted within each treatment group independently, so the pattern of missing observations in one treatment group cannot influence missing value estimations in another. For each imputation process, 25 imputations will be performed.

Subjects that withdrew from the study due to lack of efficacy will have missing values imputed, however, the WI-NRS responder status will be defined as non-responder. Subjects that used an excluded therapy to treat worsening of pruritus or PN will have data values collected after the use of the excluded therapy set to missing and subsequently imputed. These subjects will also have the WI-NRS responder status defined as non-responder.

Missing WI-NRS data will be derived for the analysis using the method of MCMC multiple imputation. The 4-point responder status will be derived from imputed WI-NRS values. Since both primary and key secondary endpoints require WI-NRS, the following steps will be followed:

- 1. Using the daily eDiary data, calculate Baseline and Week 1 through Week 10 values by averaging available values. In order to compute a week's average, a minimum of 4 values must be available for that week. The weekly average will be imputed when there are fewer than 4 values available.
- 2. From step 1, create a dataset for each treatment group, of subjects with observed values and those needing estimation by MCMC. The missing WI-NRS values in each dataset will be filled in using the MCMC method to generate 25 datasets. The resulting datasets for each treatment group will be combined into one complete dataset.

#### Syntax:

```
proc mi data=datain out=dataout seed=&seed. Nimpute=25 <options>;
  where trtpn=(TRT); /* Note TRT = [1, 2]; depending on treatment group */;
  mcmc chain=single;
  var baseline week1 week2 week3 week4 week5 week6 week7 week8 week9
      week10;
run;
```

3. From each complete dataset, the dichotomous responder rate will be determined. Each complete dataset will be analyzed as specified for the particular analysis.

The results from the analyses will be combined into a single inference using SAS® PROC MIANALYZE. In the case of the primary analysis and the secondary responder analyses, the Cochran Mantel Haenszel (CMH) statistics computed in the analyses of WI-NRS responder rates will be normalized using the Wilson-Hilferty transformation prior to combining them using SAS® PROC MIANALYZE.

A total of 2 random seeds will be needed to impute missing data. Those random seeds have been pre-specified by using a random number generator:



# 6.1.6 Interim Analyses and Data Monitoring

No interim analyses will be performed.

#### **6.1.7** Multicenter Studies

The clinical study will be conducted under a common protocol for each investigational site with the intention of pooling all data for analysis. Every effort will be made to promote consistency in study execution at each study site.

# 6.1.8 Multiple Comparisons/Multiplicity

The primary and key secondary endpoints will be analyzed. However, the statistical significance of the key secondary endpoints will only be considered should statistical significance be reached for the primary endpoint. Similarly, statistical significance within the key secondary endpoints will be considered based on a hierarchical approach, starting with the WI-NRS Week 4 responder rate followed by the WI-NRS Week 2 responder rate. If the first key secondary endpoint fails to reach statistical significance at a level of 0.05, then subsequent endpoints will not be considered statistically significant.

#### **6.1.9** Examination of Subgroups

Descriptive summaries of the primary efficacy endpoint will be created for subgroups of the Intent-to-Treat (ITT) population. Subgroups include age (< median age; >= median age), sex, ethnicity, race and Baseline WI-NRS randomization strata.

# 6.2 Disposition of Subjects

An accounting of all randomized subjects by disposition will be presented. Subjects who discontinue study drug prematurely or withdraw from the study will be summarized and listed, with a description of the reason for early termination/withdrawal.

The number of subjects included in each population will be summarized. Subjects who are excluded from a population will be summarized by the reasons for exclusion.

# 6.3 Protocol Deviations

Protocol deviations leading to exclusion from an analysis population will be tabulated. Other protocol deviations will be presented in a data listing.

#### 6.4 Data Sets Analyzed

The following analysis populations will be reviewed and approved by the Sponsor prior to unblinding the study.

# 6.4.1 Intent-to-Treat (ITT) Population

The primary efficacy population will be the ITT population, which will include all randomized subjects who were dispensed study drug. Subjects will be analyzed within the treatment group to which they are randomized.

#### **6.4.2** Safety Population

The primary safety population will be all treated subjects with at least one post-baseline assessment or a reported TEAE. For safety analyses, subjects will be classified based upon treatment received. In the case that a subject received both treatments, subjects will be summarized within the serlopitant 5 mg group.

# 6.4.3 Per Protocol Population

Additional analyses performed on the Per Protocol (PP) population will be considered supportive. The PP population will include all subjects in the safety population who complete the Week 10 evaluations without any significant protocol deviations/violations (i.e., any subject or investigator activity that could have possibly interfered with the therapeutic administration of the treatment or the precise evaluation of treatment efficacy). The PP population will include subjects in the safety population who do not meet any of the following criteria:

- Violated the inclusion/exclusion criteria;
- Received a strong CYP3A4 inhibitor (See Appendix B in the Protocol);
- Received an excluded medication which may plausibly impact the primary endpoint at Week 10 (e.g. was provided to treat pruritus or PN);
- Have not been compliant with the dosing regimen (i.e. subjects must comply with 80-120% of the expected dosage of study medication during participation in the study);
- Have not completed Week 10 visit within  $\pm 7$  days window
- Have not completed the eDiary to provide the Week 10 WI-NRS Primary Endpoint

Subjects who discontinue from the study drug due to an adverse event related to study treatment or documented lack of treatment effect, or who met protocol-defined non-responder criteria, will be included in the PP population. Prior to breaking the blind other additional criteria may be added to the lists above to accommodate for unforeseen events that occurred during the conduct of the trial that result in noteworthy study protocol deviations.

Subjects will be analyzed within the treatment group to which they are randomized.

# 6.5 Demographic and Other Baseline Characteristics

Demographic and baseline characteristics summaries will be done for the ITT, Safety, and PP populations.

Sex, race, and ethnicity will be summarized by counts and percentages. Age, height (cm), and weight (kg) will be summarized with descriptive statistics.

IGA PN-A, and IGA PN-S will be summarized by counts and percentages. WI-NRS (average result measured over the week prior to treatment) and DLQI will be summarized with descriptive statistics.

Medical histories will be coded using MedDRA, tabulated by System Organ Class and Preferred Term for the Safety population, and presented in a by-subject listing.

PN history and prior PN therapies will be presented in by-subject listings.

#### 6.6 Prior and Concomitant Medications

Prior and concomitant medications will be coded by the WHO-DDE to Anatomical Therapeutic Classification (ATC) and preferred drug name. Concomitant medications will be summarized by ATC level 2 term and preferred drug name.

A by-subject listing of all prior and concomitant medications will be presented. The associated by-subject listing will have a prior/concomitant determination that is based on the date of first dose.

#### 6.7 Analysis of Efficacy

The efficacy endpoints will be summarized within the ITT and PP populations using descriptive statistics by time point and treatment. Available results including averaged imputed values, as well as change from baseline, will be summarized for each applicable time point. The WI-NRS and change from baseline will also be presented for each study day in a by-subject listing.

For the 4- and 3-point responder rate endpoints, subjects will be considered responders if they have at least a 4- / 3-point reduction between baseline and the corresponding week. Subjects that discontinued study drug due to lack of efficacy or used an excluded medication to treat worsening of pruritus or PN will be considered non-responders.

#### 6.7.1 Primary Efficacy Analysis

The difference in the primary efficacy outcome measure (WI-NRS 4-point responder rate at Week 10) will be tested using a CMH test controlling for the 'as randomized' stratification factors. Conceptually the hypotheses being tested are:

 $H_0$ :  $P_{Placebo} \ge P_{Serlopitant}$   $H_a$ :  $P_{Placebo} < P_{Serlopitant}$ 

where  $P_{Placebo}$  is the percent of placebo responders and  $P_{Serlopitant}$  is the similar percent for serlopitant.

# 6.7.2 Key Secondary Efficacy Analysis

The WI-NRS 4-point responder rates at Week 4 and Week 2 will be analyzed using methods consistent with testing the primary endpoint.

The preceding analyses are to be conducted for the ITT and PP populations.

#### 6.7.3 Additional Secondary Efficacy Analysis

Additional secondary efficacy endpoints which may be drawn from the primary and key secondary imputations (including all WI-NRS endpoints) will be analyzed using the imputed data. Additional secondary efficacy endpoints otherwise will be analyzed using available data. P-values will be included for descriptive purposes only.

Additional secondary efficacy endpoints which are dichotomous (responder) will include analyses analogous to the primary and key secondary efficacy analyses.

Additional secondary efficacy endpoints based on change from baseline will be analyzed using an analysis of covariance (ANCOVA) model with treatment group and stratification factor as fixed effects and the baseline value as a covariate. Both least squares means and observed means will be presented.

To confirm the assumptions for the ANCOVA model (i.e., that the errors are normally distributed with equal variances), residuals will be examined using the Shapiro-Wilk test. If there is overwhelmingly strong evidence that the assumptions are not satisfied, the data will be rank-transformed prior to submitting to the ANCOVA. Results of the rank-transformed analysis then will be considered the primary analysis; however, results of the non-rank transformed analysis will also be presented.

#### 6.8 Sensitivity Analysis

#### **6.8.1** Last Observation Carried Forward

In the first set of sensitivity analyses, missing values will be imputed using LOCF. Data will be imputed using LOCF unless the subject withdrew from the study due to lack of efficacy, or the subject used an excluded therapy to treat worsening of pruritus or PN, in which case their responder status will be defined as non-responder. Each primary and key secondary endpoint will be analyzed as it was using the multiply imputed data.

# **6.8.2** Repeated Measures Analysis

The second set of sensitivity analyses will be performed on observed data.

The dichotomized primary and key secondary WI-NRS endpoints will each be analyzed with a repeated measures logistic regression model (generalized estimating equations), with the dichotomized endpoint as the dependent variable and treatment, stratification factor and visit (Weeks 1-10) as independent factors.

#### **6.8.3** Tipping Point Analysis

A sensitivity analysis for the handling of missing data for the primary efficacy endpoint will be carried out using a tipping point analysis. Specifically, a range of response rates for both groups will be explored to determine the tipping point(s) at which the combinations result in no longer reaching statistical significance.

#### 6.9 Safety Evaluation

### **6.9.1** Extent of Exposure

The extent of exposure to study drug in each treatment group will be summarized by days with exposure and total number of tablets used.

A subject will be considered compliant with the dosing regimen if the subject takes 80% to 120% of the expected number of doses while enrolled in the study. Total number of days of exposure will be computed as follows:

```
Total Exposure = Date of Last Dose – Date of First Dose + 1

Total Doses = (Date of Last Dose – Date of First Dose + 1 + 2)

– Missed Doses + Extra Doses
```

Treatment compliance will be based on the expected number of doses given the treatment period duration. The number of expected doses will be computed from the Baseline/Day 1 visit date and the Week 10 visit date. If a subject does not have a Week 10 visit, the number of expected doses will be calculated based on end of treatment period date given available information (e.g., date of last dose, last completed visit date).

```
Expected Doses = End of Treatment Period Date – Day 1 Date + 2
```

If the subject is documented as dosing on the End of Treatment Period Date, a dose will be added to the Expected Doses. To allow for the +7 day window around Week 10 that is used for defining PP population, if the number of expected doses exceeds 80, the number of expected doses will be considered 80 doses.

Percent compliance will be calculated from total number of doses and total number of expected doses as follows:

Percent Compliance = 100\*(Total Doses/Expected Doses).

Percent compliance will not be calculated for subjects who are lost to follow-up during the treatment period.

#### 6.9.2 Adverse Events

The incidence of all AEs and TEAEs will be tabulated by treatment received. These AEs will be classified by system organ class and preferred term using MedDRA. For incidence reporting, if a subject reported more than one AE that was coded to the same system organ class or preferred term, the subject will be counted only once for the specific system organ class or preferred term. An overview of AEs, which includes subject incidence of AEs, treatment-related AEs, AEs by severity, SAEs, deaths, and AEs leading to discontinuation, will be presented.

Assessment of AEs reported after study drug discontinuation will be summarized separately by treatment group. AEs during post-drug follow-up will be summarized by weekly periods and sex.

SAEs will be listed and summarized in a similar manner to AEs.

# 6.9.3 Clinical Laboratory Evaluation

Clinical safety laboratory values will be measured by a central laboratory. Summary statistics for actual values and for changes from baseline will be tabulated for laboratory results by scheduled visit.

Subjects with clinical laboratory values outside of the normal reference range at any post-baseline assessment will be summarized. Shifts from baseline laboratory values will be tabulated, with the exception of most reproductive endocrinology laboratory values.

Serum follicle-stimulating hormone, luteinizing hormone, estradiol, progesterone and antimullerian hormone will be summarized separately for women using hormonal contraception/therapies and those not using hormonal contraception/therapies.

By-subject listings of all laboratory data, as well as abnormal laboratory results, will be presented.

#### 6.9.4 Other Observations Related to Safety

#### **6.9.4.1 ECG Measurements**

Summary statistics for actual values and for changes from baseline will be tabulated for ECG parameter results by scheduled visit. The overall ECG assessment (abnormal or normal) will be summarized along with a summary of how many subjects developed a post treatment abnormal result. The study relevance of the finding (i.e. clinical significance as determined by the investigator) will be provided in a by-subject listing.

#### 6.9.4.2 Vital Signs

The observed data and change from baseline for each measurement day will be summarized with descriptive statistics, as well as provided in a by-subject listing.

#### 6.9.4.3 **Physical Exams**

Clinically significant physical exam findings will be recorded by the sites within medical history or adverse events and otherwise not summarized.

#### 6.9.4.4 Menstrual Diaries

Menstrual diary dates will be used to summarize number and duration of menses.

#### 6.9.4.5 **Hospital Anxiety and Depression Scale (HADS)**

The observed data and change from baseline for the HADS will be summarized with descriptive statistics by scheduled visit. Both the Depression and Anxiety subscales will be reported.

#### 6.9.4.6 **Epworth Sleepiness Scale (ESS)**

The observed data and change from baseline for the ESS will be summarized with descriptive statistics by scheduled visit.

#### 6.10 **Pharmacokinetic Analysis**

The plasma concentrations of serlopitant and metabolites will be summarized using descriptive statistics.

By-subject listings of the plasma concentrations of serlopitant and metabolites will be presented.

#### **DETERMINATION OF SAMPLE SIZE**

This study will use a 5% two-sided alpha level. While the alpha level is two-sided, clinically relevant results require a serlopitant benefit.

The target sample size of 280 randomized and dosed subjects (140 per group) has been determined based upon a 1:1 allocation of subjects to treatment groups and a 5% alpha level. Completed Phase 2 studies indicate that placebo responder rates vary between \(\frac{co}{\circ}\)% and \(\frac{co}{\circ}\)% and serlopitant rates between % and %. A sample size of 280 subjects provides >90% power assuming a placebo responder rate of "" and serlopitant rate of ".

The sample size calculations have been performed in PASS 13 ("PASS 13 Power Analysis and Sample Size Software" 2014) and use a Chi-Squared test. The primary analysis will control for the stratification factors. It is expected that this unstratified power estimate will under-estimate

the true power as it does not take the variance reduction resulting from stratification into account (Matts 1988).

#### 8. CHANGES IN THE PLANNED ANALYSES

No changes to planned analyses.

#### 9. REFERENCES

- Jorizzo JL, Gatti S, Smith EB. Prurigo: a clinical review. J Am Acad Dermatol. 1981;4(6): 723-728.
- Matts JP LJ. Properties of permuted-block randomization in clinical trials. *Control ClinTrials*. 1988;9(4):327-344.
- PASS 13 Power Analysis and Sample Size Software [computer program]. Kaysville, Utah, USA, ncss.com/software/pass.: NCSS, LLC; 2014.
- Zeidler C, Ständer S. The pathogenesis of prurigo nodularis--'Super-Itch' in exploration. Eu J Pain. 2016;20(1):37-40.

Statistical Analysis Plan for Menlo Therapeutics Inc. Protocol Number: MTI-106 16 December 2019

Page 20

# 10. INDEX OF PLANNED END-OF-TEXT TABLES AND FIGURES

| Table 14.0.1: Summary of Subject Completion/Discontinuation (Randomized Subjects) | 26 |
|---|---|
| Table 14.0.2: Summary of Subjects Excluded from Analyses (Randomized Subjects) | 27 |
| Table 14.0.3: Summary of Subject Visit Attendance (Randomized Subjects) | 28 |
| Table 14.1.1.1: Summary of Subject Demographics (Intent-to-Treat Population) | 29 |
| Table 14.1.1.2: Summary of Subject Demographics (Per-Protocol Population) | 30 |
| Table 14.1.1.3: Summary of Subject Demographics (Safety Population) | 30 |
| Table 14.1.2.1: Subject Baseline Characteristics (Intent-to-Treat Population) | 31 |
| Table 14.1.2.2: Subject Baseline Characteristics (Per-Protocol Population) | 32 |
| Table 14.1.2.3: Subject Baseline Characteristics (Safety Population) | 32 |
| Table 14.1.3: Summary of Medical History by MedDRA System Organ Class and Preferred Term (Intent-to-Treat Population) | 33 |
| Table 14.1.4: Summary of Concomitant Medications by ATC Level 2 Term and Preferred Drug Name (Intent-to-Treat Population) | |
| Table 14.2.1.1: Analysis of the Primary Efficacy Endpoint: Worst-Itch Numeric Rating Scale (WI-NRS) 4-Point Responder at Week 10 (Intent-to-Treat Population) | 35 |
| Table 14.2.1.2: Analysis of the Primary Efficacy Endpoint: Worst-Itch Numeric Rating Scale (WI-NRS) 4-Point Responder at Week 10 (Per-Protocol Population). | 35 |
| Table 14.2.1.3: Sensitivity Analyses of the Primary Efficacy Endpoint: Worst-Itch Numeric Rating Scale (WI-NRS) 4-Point Responder at Week 10 (Intent-to-Treat Population) | |
| Figure 14.2.1.4: Sensitivity Tipping-Point Analyses of the Primary Efficacy Endpoint: Worst-<br>Itch Numeric Rating Scale (WI-NRS) 4-Point Responder at Week 10<br>(Intent-to-Treat Population) | |
| Table 14.2.1.4: Subgroup Summaries of Primary Efficacy Endpoint: Worst-Itch Numeric Rating Scale (WI-NRS) 4-Point Responder at Week 10 (Intent-to-Treat Population) | Č |
| Table 14.2.2.1: Analysis of Key Secondary Efficacy Endpoints (Intent-to-Treat Population) | 41 |
| Table 14.2.2.2: Analysis of Key Secondary Efficacy Endpoints (Per-Protocol Population) | 41 |
| Table 14.2.2.3: Sensitivity Analyses of Key Secondary Efficacy Endpoints (Intent-to-Treat Population) | 42 |
| Table 14.2.3.1: Analysis of Additional Secondary Efficacy Endpoints (Intent-to-Treat Population) | 44 |
| Table 14.2.3.2: Analysis of Additional Secondary Efficacy Endpoints (Per-Protocol Population) | 50 |

| Table 14.2.4.1: Summary of Worst Itch Numeric Rating Scale (WI-NRS) (Intent-to-Treat Population) |
|---|
| Table 14.2.4.2: Summary of Worst Itch Numeric Rating Scale (WI-NRS) (Per-Protocol Population) |
| Table 14.2.4.3: Summary of Worst Itch Numeric Rating Scale (WI-NRS) – Observed Data with Follow-up (Intent-to-Treat Population with Observed Week 10 Data) |
| Table 14.2.5.1.1: Summary of Dermatology Life Quality Index (DLQI) (Intent-to-Treat Population) |
| Table 14.2.5.1.2: Summary of Dermatology Life Quality Index (DLQI) (Per-Protocol Population) |
| Table 14.2.5.2.1: Summary of Dermatology Life Quality Index (DLQI) Individual Questions (Intent-to-Treat Population) |
| Table 14.2.5.2.2: Summary of Dermatology Life Quality Index (DLQI) – Individual Questions (Per-Protocol Population) |
| Table 14.2.6.1: Summary of Investigator's Global Assessment of Prurigo Nodularis Activity (IGA PN-A) (Intent-to-Treat Population) |
| Table 14.2.6.2: Summary of Investigator's Global Assessment of Prurigo Nodularis Activity (IGA PN-A) (Per-Protocol Population) |
| Table 14.2.7.1: Summary of Investigator's Global Assessment of Prurigo Nodularis Stage (IGA PN-S) (Intent-to-Treat Population) |
| Table 14.2.7.2: Summary of Investigator's Global Assessment of Prurigo Nodularis Stage (IGA PN-S) (Per-Protocol Population) |
| Table 14.3.0.1: Summary of Extent of Exposure (Intent-to-Treat Population) |
| Table 14.3.0.2: Summary of Extent of Exposure (Per-Protocol Population) |
| Table 14.3.0.3: Summary of Extent of Exposure (Safety Population) |
| Table 14.3.1.1.1: Overall Summary of Treatment-Emergent Adverse Events (TEAEs) (Safety Population) |
| Table 14.3.1.1.2: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.1.3: Summary of Treatment-Emergent Adverse Events (TEAEs) Leading to Discontinuation of Study Drug (Safety Population)80 |
| Table 14.3.1.1.4: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population) |
| Table 14.3.1.1.5: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug (Safety Population)82 |
| Table 14.3.1.2.1.1: Overall Summary of Post-Drug Adverse Event (AEs) (Safety Population)83 |

| Table 14.3.1.2.1.2: Overall Summary of Post-Drug Adverse Events (AEs) Occurring 1-7 Days Post Last Dose (Safety Population) |
|---|
| Table 14.3.1.2.1.3: Overall Summary of Post-Drug Adverse Events (AEs) Occurring 8-14 Days Post Last Dose (Safety Population) |
| Table 14.3.1.2.1.4: Overall Summary of Post-Drug Adverse Events (AEs) Occurring 15-21 Days Post Last Dose (Safety Population) |
| Table 14.3.1.2.1.5: Overall Summary of Post-Drug Adverse Events (AEs) Occurring 22-28 Days Post Last Dose (Safety Population) |
| Table 14.3.1.2.1.6: Overall Summary of Post-Drug Adverse Events (AEs) Occurring 29-35 Days Post Last Dose (Safety Population) |
| Table 14.3.1.2.2.1: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.2.2.2: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 1-7 Days Post Last Dose by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.2.2.3: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 8-14 Days Post Last Dose by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.2.2.4: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 15-21 Days Post Last Dose by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.2.2.5: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 22-28 Days Post Last Dose by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.2.2.6: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 29-35 Days Post Last Dose by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.2.3.1: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) by Severity (Safety Population) |
| Table 14.3.1.2.3.2: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 1-7 Days Post Last Dose by Severity (Safety Population)90 |
| Table 14.3.1.2.3.3: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 8-14 Days Post Last Dose by Severity (Safety Population)91 |
| Table 14.3.1.2.3.4: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 15-21 Days Post Last Dose by Severity (Safety Population)91 |
| Table 14.3.1.2.3.5: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 22-28 Days Post Last Dose by Severity (Safety Population)91 |
| Table 14.3.1.2.3.6: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 29-35 Days Post Last Dose by Severity (Safety Population)91 |

| Table 14.3.1.2.4.1: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) by Relationship to Study Drug (Safety Population) |
|---|
| Table 14.3.1.2.4.2: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 1-7 Days Post Last Dose by Relationship to Study Drug (Safety Population) 93 |
| Table 14.3.1.2.4.3: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 8-14 Days Post Last Dose by Relationship to Study Drug (Safety Population) |
| Table 14.3.1.2.4.4: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 15-21 Days Post Last Dose by Relationship to Study Drug (Safety Population) |
| Table 14.3.1.2.4.5: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 22-28 Days Post Last Dose by Relationship to Study Drug (Safety Population) |
| Table 14.3.1.2.4.6: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 29-35 Days Post Last Dose by Relationship to Study Drug (Safety Population) |
| Table 14.3.1.3.1: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.3.2: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population)96 |
| Table 14.3.1.3.3: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug (Safety Population)97 |
| Table 14.3.1.4.1.1: Summary of Hematology Laboratory Results (Safety Population)98 |
| Table 14.3.1.4.1.2: Shift Summary of Hematology Laboratory Results (Safety Population)99 |
| Table 14.3.1.4.2.1: Summary of Chemistry Laboratory Results (Safety Population)100 |
| Table 14.3.1.4.2.2: Shift Summary of Chemistry Laboratory Results (Safety Population)103 |
| Table 14.3.1.4.3.1.1: Summary of Endocrine/Reproductive Endocrine Laboratory Results (Safety Population) |
| Table 14.3.1.4.3.1.2: Summary of Reproductive Endocrine Laboratory Results (Safety Population – Females Using Hormonal Contraception/Therapy) |
| Table 14.3.1.4.3.1.3: Summary of Reproductive Endocrine Laboratory Results (Safety Population – Females Not Using Hormonal Contraception/Therapy) |
| Table 14.3.1.4.3.2: Shift Summary of Endocrine/Reproductive Endocrine Laboratory Results (Safety Population) |

| Table 14.3.1.5.1.1: Summary of Treatment-Emergent Electrocardiogram (ECG) Parameter Abnormalities (Safety Population) | .106 |
|---|---|
| Table 14.3.1.5.1.2: Summary of Electrocardiogram Parameters (Safety Population) | .108 |
| Table 14.3.1.5.1.3: Shift Summary of Overall Electrocardiogram (ECG) Assessments (Safety Population) | |
| Table 14.3.1.6.1: Summary of Vital Signs (Safety Population) | .111 |
| Table 14.3.1.7.1: Summary of Hospital Anxiety and Depression Scale (HADS) (Safety Population) | .112 |
| Table 14.3.1.8.1: Summary of Epworth Sleepiness Scale (ESS) (Safety Population) | .113 |
| Table 14.3.1.9: Summary of Pharmacokinetic Concentrations (Safety Population) | .114 |
| Table 14.3.1.10: Summary of Menstrual Cycles (Safety Population) | .115 |

Table 14.0.1: Summary of Subject Completion/Discontinuation (Randomized Subjects)

| | Placebo | Serlopitant 5 mg |
|---|---|---|
| | (N=xxx) | (N=xxx) |
| Completed Treatment | | · |
| Yes | xx ( xx.x%) | xx ( xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) |
| Reason for Discontinuation from Treatment | | |
| Adverse Event | xx ( xx.x%) | xx ( xx.x%) |
| Lack of Efficacy | xx ( xx.x%) | xx ( xx.x%) |
| Pregnancy | xx ( xx.x%) | xx ( xx.x%) |
| Investigator Decision | xx ( xx.x%) | xx ( xx.x%) |
| Withdrawal by Subject from Treatment | xx ( xx.x%) | xx ( xx.x%) |
| Protocol Deviation | xx ( xx.x%) | xx ( xx.x%) |
| Sponsor Decision | xx ( xx.x%) | xx ( xx.x%) |
| Other | xx ( xx.x%) | xx ( xx.x%) |
| Completed Follow-up | | |
| Yes | xx (xx.x%) | xx ( xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) |
| Reason for Discontinuation from Follow-up | | |
| Withdrawal by Subject from Study | xx (xx.x%) | xx ( xx.x%) |
| Lost to Follow-up | xx ( xx.x%) | xx ( xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) |

Table 14.0.2: Summary of Subjects Excluded from Analyses (Randomized Subjects)

| | Placebo | Serlopitant 5 mg |
|--------------------------------------------|-------------|------------------|
| _ | (N=xxx) | (N=xxx) |
| Intent-to-Treat Population | | |
| Number of Subjects Included | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded | xx ( xx.x%) | xx ( xx.x%) |
| Reason for Exclusion | | |
| Not Dispensed Study Drug | xx ( xx.x%) | xx ( xx.x%) |
| <b>Safety Population</b> | | |
| Number of Subjects Included | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded | xx ( xx.x%) | xx ( xx.x%) |
| Reason for Exclusion | | |
| No Evidence of Subject Dosing | xx ( xx.x%) | xx ( xx.x%) |
| No Post-Baseline Assessment/TEAE | xx ( xx.x%) | xx ( xx.x%) |
| Per-Protocol Population | | |
| Number of Subjects Included | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded | xx ( xx.x%) | xx ( xx.x%) |
| Reason for Exclusion | | |
| No Evidence of Subject Dosing | xx ( xx.x%) | xx ( xx.x%) |
| No Post-Baseline Assessment/TEAE | xx ( xx.x%) | xx ( xx.x%) |
| Violated the Inclusion/Exclusion Criteria | xx ( xx.x%) | xx ( xx.x%) |
| Received a Strong CYP3A4 Inhibitor | xx ( xx.x%) | xx ( xx.x%) |
| Received an Excluded Medication | xx ( xx.x%) | xx ( xx.x%) |
| Was not Compliant with the Dosing Regimen | xx ( xx.x%) | xx ( xx.x%) |
| Week 10 WI-NRS Data Not Available | xx ( xx.x%) | xx ( xx.x%) |
| Did not Attend the Week 10 Visit | xx ( xx.x%) | xx ( xx.x%) |
| Week 10 Visit not within +/- 7 days Window | xx ( xx.x%) | xx ( xx.x%) |

Note: TEAE = Treatment Emergent Adverse Event; WI-NRS=Worst-Itch Numeric Rating Scale

Table 14.0.3: Summary of Subject Visit Attendance (Randomized Subjects)

| | Placebo | Serlopitant 5 mg |
|--------------------|-------------|------------------|
| Subjects Attending | (N=xxx) | (N=xxx) |
| Screening | xx ( xx.x%) | xx ( xx.x%) |
| Baseline | xx (xx.x%) | xx ( xx.x%) |
| Week 2 | xx (xx.x%) | xx ( xx.x%) |
| Week 4 | xx ( xx.x%) | xx ( xx.x%) |
| Week 6 | XX (XX.X%) | XX (XX.X%) |
| Week 10 | xx ( xx.x%) | xx ( xx.x%) |
| 3-Week Follow-up | xx ( xx.x%) | xx ( xx.x%) |
| 5-Week Follow-up | xx ( xx.x%) | XX (XX.X%) |

Table 14.1.1.1: Summary of Subject Demographics (Intent-to-Treat Population) 

| | Placebo | Serlopitant 5 mg | Total |
|---|---|---|---|
| _ | (N=xxx) | N=xxx | (N=xxx) |
| Age (years) | | | |
| n | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Sex | | | |
| n | xxx | XXX | XXX |
| Male | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Female | XX (XX.X%) | xx ( xx.x%) | xx ( xx.x%) |
| Ethnicity | | | |
| n | XXX | XXX | XXX |
| Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Race | | | |
| n | XXX | XXX | XXX |
| American Indian or Alaska Native | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Asian | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Black or African American | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| White | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Multiple/Other | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Table 14.1.1.1: Summary of Subject Demographics (Intent-to-Treat Population) 

| | Placebo | Serlopitant 5 mg | Total<br>(N=xxx) |
|--------------|------------|------------------|------------------|
| | (N=xxx) | N=xxx | |
| Height (cm) | | | |
| n | XXX | XXX | XXX |
| Mean | XXX.X | XXX.X | XXX.X |
| SD | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.X | XXX.X | XXX.X |
| Min. to Max. | xxx to xxx | xxx to xxx | xxx to xxx |
| Weight (kg) | | | |
| n | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xxx | xx to xxx | xx to xxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.1.1.1 for the following:

Table 14.1.1.2: Summary of Subject Demographics (Per-Protocol Population)

Table 14.1.1.3: Summary of Subject Demographics (Safety Population)

Table 14.1.2.1: Subject Baseline Characteristics (Intent-to-Treat Population) 

| | Placebo | Serlopitant 5 mg | Total |
|---|---|---|---|
| _ | (N=xxx) | (N=xxx) | N=xxx |
| Baseline WI-NRS (1-Week Average Prior to | | | |
| Baseline) | | | |
| n | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Investigator's Global Assessment of Prurigo | | | |
| Nodularis Activity | | | |
| n | XXX | XXX | XXX |
| Grade 0 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Investigator's Global Assessment of Prurigo | | | |
| Nodularis Stage | | | |
| n | XXX | XXX | XXX |
| Grade 0 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Table 14.1.2.1: Subject Baseline Characteristics (Intent-to-Treat Population) 

| | Placebo (N=xxx) | Serlopitant 5 mg<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Dermatology Life Quality Index | | | |
| n | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.1.2.1 for the following:

Table 14.1.2.2: Subject Baseline Characteristics (Per-Protocol Population)

Table 14.1.2.3: Subject Baseline Characteristics (Safety Population)

Table 14.1.3: Summary of Medical History by MedDRA System Organ Class and Preferred Term (Intent-to-Treat Population)

| System Organ Class <sup>a</sup> | Placebo | Serlopitant 5 mg | Total |
|---|---|---|---|
| Preferred Term | (N=xxx) | (N=xxx) | (N=xxx) |
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more medical histories that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Note: MedDRA Version 21.1.

Table 14.1.4: Summary of Concomitant Medications by ATC Level 2 Term and Preferred Drug Name (Intent-to-Treat Population)


| ATC Level 2 Term <sup>a</sup> | Placebo | Serlopitant 5 mg | Total |
|-------------------------------|-------------|------------------|-------------|
| Preferred Drug Name | (N=xxx) | (N=xxx) | (N=xxx) |
| ATC Level 2 Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Drug Name | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ATC Level 2 Term | | | |
| Preferred Drug Name | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more concomitant medications that map to the WHO-DDE. At each level of summarization (ATC Level 2 Term or Standard Medication Name) subjects are counted once.

Note: WHO Drug Dictionary, Version September 1, 2018.

Table 14.2.1.1: Analysis of the Primary Efficacy Endpoint: Worst-Itch Numeric Rating Scale (WI-NRS) 4-Point Responder at Week 10 (Intent-to-Treat Population)

| | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) | P-value <sup>a</sup> |
|---|---|---|---|
| At Least 4-Point Reduction from Baseline in | · | | |
| Weekly Average WI-NRS at Week 10 | | | |
| Success | xx.xx% | XX.XX <sup>0</sup> / <sub>0</sub> | X.XXX |
| Failure | XX.XX <sup>0</sup> / <sub>0</sub> | XX.XX <sup>0</sup> / <sub>0</sub> | |

<sup>&</sup>lt;sup>a</sup> P-value from a Cochran Mantel Haenszel (CMH) test stratified by Baseline WI-NRS used for randomization stratification. Value has been adjusted for multiple imputation.

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics represent average values, obtained by averaging the summary statistics generated from each imputed dataset.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.1.1 for the following:

Table 14.2.1.2: Analysis of the Primary Efficacy Endpoint: Worst-Itch Numeric Rating Scale (WI-NRS) 4-Point Responder at Week 10 (Per-Protocol Population)
Table 14.2.1.3: Sensitivity Analyses of the Primary Efficacy Endpoint: Worst-Itch Numeric Rating Scale (WI-NRS) 4-Point Responder at Week 10 (Intent-to-Treat Population)

| | Placebo | Serlopitant 5 mg | |
|---|---|---|---|
| <u> </u> | (N=xxx) | (N=xxx) | P-value |
| Missing Values Imputed using Last | | | |
| <b>Observation Carried Forward (LOCF)</b> | | | |
| At Least 4-Point Reduction from Baseline in | | | |
| Weekly Average WI-NRS at Week 10 | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | X.XXX <sup>a</sup> |
| Failure | XX ( XX.X%) | xx ( xx.x%) | |
| Repeated Measures Analysis on Observed | | | |
| Data | | | |
| At Least 4-Point Reduction from Baseline in | | | |
| Weekly Average WI-NRS at Week 10 | | | |
| Success | xx.xx% | XX.XX <sup>0</sup> / <sub>0</sub> | $x.xxx^b$ |
| Failure | XX.XX <sup>0</sup> / <sub>0</sub> | xx.xx% | |

<sup>&</sup>lt;sup>a</sup> P-value from a Cochran Mantel Haenszel (CMH) test stratified by Baseline WI-NRS randomization stratification.

<sup>&</sup>lt;sup>b</sup> P-value from a repeated measures logistic regression with factors of treatment group, randomization stratification, visit and treatment group by visit interaction.

Figure 14.2.1.4: Sensitivity Tipping-Point Analyses of the Primary Efficacy Endpoint: Worst-Itch Numeric Rating Scale (WI-NRS)

4-Point Responder at Week 10

(Intent-to-Treat Population)



Note: The horizontal and vertical axes indicate the potential number of successes among subjects with missing data in each treatment group.

Each plotted point indicates the number of imputed successes in each treatment group that results in p-value greater than 0.05.

The red lines represent average number of imputed successes from the primary analysis using multiple imputation (MCMC) to impute missing values.

Table 14.2.1.4: Subgroup Summaries of Primary Efficacy Endpoint: Worst-Itch Numeric Rating Scale (WI-NRS) 4-Point Responder at Week 10 (Intent-to-Treat Population)


| Sex | | Male | Fe | emale |
|---|---|---|---|---|
| | Placebo | Serlopitant 5mg | Placebo | Serlopitant 5mg |
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| At Least 4-Point Reduction from Baseline in | | | | |
| Weekly Average WI-NRS at Week 10 | | | | |
| Success | xx.xx% | xx.xx% | xx.xx% | xx.xx% |
| Failure | XX.XX <sup>0</sup> / <sub>0</sub> | XX.XX <sup>0</sup> /o | XX.XX <sup>0</sup> / <sub>0</sub> | xx.xx% |
| Age | Age < Me | edian Age (xx) | Age >= Me | edian Age (xx) |
| | Placebo | Serlopitant 5mg | Placebo | Serlopitant 5mg |
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| At Least 4-Point Reduction from Baseline in | | | ` ' | |
| Weekly Average WI-NRS at Week 10 | | | | |
| Success | xx.xx% | xx.xx% | xx.xx% | xx.xx% |
| Failure | XX.XX <sup>0</sup> / <sub>0</sub> | XX.XX <sup>0</sup> / <sub>0</sub> | xx.xx% | XX.XX <sup>0</sup> / <sub>0</sub> |
| WI-NRS Randomization Strata | WI-NRS | WI-NRS of 6.5 to <9 | | S of 9 to 10 |
| | Placebo | Serlopitant 5mg | Placebo | Serlopitant 5mg |
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| At Least 4-Point Reduction from Baseline in | <del>-</del> | | * | |
| Weekly Average WI-NRS at Week 10 | | | | |
| Success | xx.xx% | xx.xx% | xx.xx% | xx.xx% |
| Failure | xx.xx% | XX.XX% | xx.xx <sup>0</sup> / <sub>0</sub> | xx.xx <sup>0</sup> / <sub>0</sub> |

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics represent average values, obtained by averaging the summary statistics generated from each imputed dataset.

Table 14.2.1.4: Subgroup Summary of Primary Efficacy Endpoint: Worst-Itch Numeric Rating Scale (WI-NRS) 4-Point Responder at Week 10 (Intent-to-Treat Population)


| Ethnicity | Hispan | ic or Latino | Not Hispa | anic or Latino |
|---|---|---|---|---|
| · | Placebo | Serlopitant 5mg | Placebo | Serlopitant 5mg |
| | N=xxx | (N=xxx) | (N=xxx) | (N=xxx) |
| At Least 4-Point Reduction from Baseline in | • | | | - |
| Weekly Average WI-NRS at Week 10 | | | | |
| Success | xx.xx% | XX.XX% | XX.XX <sup>0</sup> / <sub>0</sub> | xx.xx% |
| Failure | XX.XX <sup>0</sup> / <sub>0</sub> | XX.XX <sup>0</sup> / <sub>0</sub> | xx.xx% | XX.XX <sup>0</sup> / <sub>0</sub> |
| Race | Black or A | frican American | 7 | White |
| | Placebo | Serlopitant 5mg | Placebo | Serlopitant 5mg |
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| At Least 4-Point Reduction from Baseline in | | | ` ' | |
| Weekly Average WI-NRS at Week 10 | | | | |
| Success | XX.XX <sup>0</sup> / <sub>0</sub> | XX.XX <sup>0</sup> / <sub>0</sub> | xx.xx% | XX.XX <sup>0</sup> / <sub>0</sub> |
| Failure | xx.xx% | xx.xx% | xx.xx% | XX.XX <sup>0</sup> / <sub>0</sub> |
| Race (continued) | American India | an or Alaska Native | A | Asian |
| , | Placebo | Serlopitant 5mg | Placebo | Serlopitant 5mg |
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| At Least 4-Point Reduction from Baseline in | · · · · · · | | * | - <del> </del> |
| Weekly Average WI-NRS at Week 10 | | | | |
| Success | xx.xx% | XX.XX <sup>0</sup> /o | xx.xx% | xx.xx% |
| Failure | xx.xx% | XX.XX <sup>0</sup> / <sub>0</sub> | xx.xx% | xx.xx% |

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics represent average values, obtained by averaging the summary statistics generated from each imputed dataset.

Table 14.2.1.4: Subgroup Summary of Primary Efficacy Endpoint: Worst-Itch Numeric Rating Scale (WI-NRS) 4-Point Responder at Week 10 (Intent-to-Treat Population)


| Race (continued) | Native Hawaiian or Other Pacific Islander | | Multiple/Other | |
|---|---|---|---|---|
| | Placebo | Serlopitant 5mg | Placebo | Serlopitant 5mg |
| | N=xxx | (N=xxx) | (N=xxx) | (N=xxx) |
| At Least 4-Point Reduction from Baseline in | | | | |
| Weekly Average WI-NRS at Week 10 | | | | |
| Success | XX.XX <sup>0</sup> / <sub>0</sub> | xx.xx% | xx.xx% | xx.xx% |
| Failure | XX.XX <sup>0</sup> / <sub>0</sub> | XX.XX <sup>0</sup> /o | XX.XX <sup>0</sup> / <sub>0</sub> | $XX.XX^{0}/_{0}$ |

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics represent average values, obtained by averaging the summary statistics generated from each imputed dataset.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.2.1: Analysis of Key Secondary Efficacy Endpoints (Intent-to-Treat Population)

| | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) | P-value <sup>a</sup> |
|---|---|---|---|
| At Least 4-Point Reduction from Baseline in | | | |
| Weekly Average Worst Itch Numeric Rating | | | |
| Scale (WI-NRS) at Week 4 | | | |
| Success | XX.XX <sup>0</sup> / <sub>0</sub> | XX.XX% | X.XXX |
| Failure | xx.xx% | XX.XX% | |
| At Least 4-Point Reduction from Baseline in<br>Weekly Average Worst Itch Numeric Rating<br>Scale (WI-NRS) at Week 2<br>Success | xx.xx% | xx.xx% | V V V V |
| | | | X.XXX |
| Failure | XX.XX <sup>0</sup> / <sub>0</sub> | xx.xx% | |

<sup>&</sup>lt;sup>a</sup> P-value from a Cochran Mantel Haenszel (CMH) test stratified by Baseline WI-NRS used for randomization stratification. Value has been adjusted for multiple imputation.

Note: Multiple imputation (MCMC) used to impute missing values. Change calculated as post-baseline – baseline.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.2.1 for the following:

Table 14.2.2.2: Analysis of Key Secondary Efficacy Endpoints (Per-Protocol Population)

Table 14.2.2.3: Sensitivity Analyses of Key Secondary Efficacy Endpoints (Intent-to-Treat Population) 

| Missing Values Imputed using Last Observation Carried Forward (LOCF) At Least 4-Point Reduction from Baseline in Weekly Average Worst Itch Numeric Rating Scale (WI-NRS) at Week 4 | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) | P-value |
|---|---|---|---|
| Success | xx ( xx.x%) | xx ( xx.x%) | X.XXX <sup>a</sup> |
| Failure | xx ( xx.x%) | xx ( xx.x%) | |
| At Least 4-Point Reduction from Baseline in<br>Weekly Average Worst Itch Numeric Rating<br>Scale (WI-NRS) at Week 2<br>Success | xx ( xx.x%) | xx ( xx.x%) | x.xxx <sup>a</sup> |
| Failure | xx ( xx.x%) | xx ( xx.x%) | |

P-value from a Cochran Mantel Haenszel (CMH) test stratified by Baseline WI-NRS used for randomization stratification.
 P-value from a repeated measures logistic regression with factors of treatment group, randomization stratification, visit and treatment group by visit interaction.

Table 14.2.2.3: Sensitivity Analyses of Key Secondary Efficacy Endpoints (Intent-to-Treat Population) 

| Repeated Measures Analysis on Observed Data At Least 4-Point Reduction from Baseline in Weekly Average Worst Itch Numeric Rating Scale (WI-NRS) at Week 4 | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) | P-value |
|---|---|---|---|
| Success<br>Failure | xx.xx%<br>xx.xx% | xx.xx%<br>xx.xx% | $x.xxx^b$ |
| At Least 4-Point Reduction from Baseline in<br>Weekly Average Worst Itch Numeric Rating<br>Scale (WI-NRS) at Week 2<br>Success<br>Failure | xx.xx%<br>xx.xx% | xx.xx%<br>xx.xx% | x.xxx <sup>b</sup> |

P-value from a Cochran Mantel Haenszel (CMH) test stratified by Baseline WI-NRS used for randomization stratification.
 P-value from a repeated measures logistic regression with factors of treatment group, randomization stratification, visit and treatment group by visit interaction.

Table 14.2.3.1: Analysis of Additional Secondary Efficacy Endpoints (Intent-to-Treat Population)


| | Placebo (N=xxx) | Serlopitant 5 mg (N=xxx) | Normality<br>P-Value | Treatment<br>P-Value |
|---|---|---|---|---|
| Weekly Average Worst Itch Numeric Rating | · | | | |
| Scale (WI-NRS) – Absolute Change from | | | | |
| Baseline to Week 2 | | | | |
| LS Mean <sup>a</sup> | x.xx | x.xx | $x.xxx^b$ | x.xxx <sup>a</sup> |
| LS SD <sup>a</sup> | x.xxx | x.xxx | | x.xxx <sup>c</sup> |
| Median <sup>d</sup> | X.XX | x.xx | | |
| Min. to Max. <sup>d</sup> | x.x to x.x | x.x to x.x | | |
| Weekly Average Worst Itch Numeric Rating | | | | |
| Scale (WI-NRS) – Absolute Change from | | | | |
| Baseline to Week 4 | | | | |
| LS Mean <sup>a</sup> | x.xx | x.xx | $x.xxx^b$ | x.xxx <sup>a</sup> |
| LS SD <sup>a</sup> | x.xxx | x.xxx | | x.xxx <sup>c</sup> |
| Median <sup>d</sup> | x.xx | x.xx | | |
| Min. to Max.d | x.x to x.x | x.x to x.x | | |

<sup>&</sup>lt;sup>a</sup> P-values, least squares means (LS Mean) and standard deviations (LS SD) from an analysis of covariance (ANCOVA) with treatment group and stratification factor as fixed effects, and baseline value as a covariate. Values have been adjusted for multiple imputation.

<sup>&</sup>lt;sup>b</sup> P-value from a Shapiro-Wilk test for normality. Average p-value across imputations is presented.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance (ANCOVA) with treatment group and stratification factor as fixed effects, and baseline value as a covariate. Value has been adjusted for multiple imputation.

d Median, minimum and maximum represent average values, obtained from averaging the summary statistics generated from each imputed dataset. Note: Multiple imputation (MCMC) used to impute missing values. Change calculated as post-baseline – baseline. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.3.1: Analysis of Additional Secondary Efficacy Endpoints (Intent-to-Treat Population) 

| | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) | Normality<br>P-Value | Treatment<br>P-Value |
|---|---|---|---|---|
| Weekly Average Worst Itch Numeric Rating | <del></del> | | | |
| Scale (WI-NRS) – Absolute Change from | | | | |
| Baseline to Week 6 | | | | |
| LS Mean <sup>a</sup> | x.xx | X.XX | $x.xxx^b$ | x.xxx <sup>a</sup> |
| LS SD <sup>a</sup> | x.xxx | x.xxx | | x.xxx <sup>c</sup> |
| Median <sup>d</sup> | X.XX | x.xx | | |
| Min. to Max. <sup>d</sup> | x.x to x.x | x.x to x.x | | |
| Weekly Average Worst Itch Numeric Rating | | | | |
| Scale (WI-NRS) – Absolute Change from | | | | |
| Baseline to Week 10 | | | | |
| LS Mean <sup>a</sup> | x.xx | x.xx | $x.xxx^b$ | x.xxx <sup>a</sup> |
| LS SD <sup>a</sup> | x.xxx | x.xxx | | x.xxx <sup>c</sup> |
| Median <sup>d</sup> | x.xx | x.xx | | |
| Min. to Max.d | x.x to x.x | x.x to x.x | | |

<sup>&</sup>lt;sup>a</sup> P-values, least squares means (LS Mean) and standard deviations (LS SD) from an analysis of covariance (ANCOVA) with treatment group and stratification factor as fixed effects, and baseline value as a covariate. Values have been adjusted for multiple imputation.

Note: Multiple imputation (MCMC) used to impute missing values. Change calculated as post-baseline – baseline.

<sup>&</sup>lt;sup>b</sup> P-value from a Shapiro-Wilk test for normality. Average p-value across imputations is presented.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance (ANCOVA) with treatment group and stratification factor as fixed effects, and baseline value as a covariate. Value has been adjusted for multiple imputation.

d Median, minimum and maximum represent average values, obtained from averaging the summary statistics generated from each imputed dataset.

<sup>&</sup>lt;sup>e</sup> P-value from a Cochran Mantel Haenszel (CMH) test stratified by Baseline WI-NRS used for randomization stratification. Value has been adjusted for multiple imputation.

Table 14.2.3.1: Analysis of Additional Secondary Efficacy Endpoints (Intent-to-Treat Population)


| | Placebo<br>(N=xxx) | Serlopitant 5 mg<br>(N=xxx) | Normality<br>P-Value | Treatment<br>P-Value |
|---|---|---|---|---|
| At Least 3-Point Reduction from Baseline in Weekly Average Worst Itch Numeric Rating | | | | |
| Scale (WI-NRS) at Week 2 | | | | |
| Success | XX.XX <sup>0</sup> / <sub>0</sub> | XX.XX <sup>0</sup> /o | N/A | x.xxx <sup>a</sup> |
| Failure | XX.XX <sup>0</sup> / <sub>0</sub> | XX.XX <sup>0</sup> / <sub>0</sub> | | |
| At Least 3-Point Reduction from Baseline in<br>Weekly Average Worst Itch Numeric Rating<br>Scale (WI-NRS) at Week 4 | | | | |
| Success | XX.XX <sup>0</sup> / <sub>0</sub> | xx.xx% | N/A | x.xxx <sup>a</sup> |
| Failure | XX.XX <sup>0</sup> / <sub>0</sub> | XX.XX <sup>0</sup> / <sub>0</sub> | | |
| At Least 3-Point Reduction from Baseline in<br>Weekly Average Worst Itch Numeric Rating<br>Scale (WI-NRS) at Week 10 | | | | |
| Success | XX.XX% | XX.XX% | N/A | x.xxx <sup>a</sup> |
| Failure | XX.XX% | XX.XX% | | |

<sup>&</sup>lt;sup>a</sup> P-value from a Cochran Mantel Haenszel (CMH) test stratified by Baseline WI-NRS used for randomization stratification. Value has been adjusted for multiple imputation.

Note: Multiple imputation (MCMC) used to impute missing values.

Table 14.2.3.1: Analysis of Additional Secondary Efficacy Endpoints (Intent-to-Treat Population)


| | Placebo (N=xxx) | Serlopitant 5 mg (N=xxx) | Normality<br>P-Value | Treatment P-Value |
|---|---|---|---|---|
| Investigator's Global Assessment of Prurigo | (IV AAA) | (IV AAA) | 1 value | 1 value |
| Nodularis Activity (IGA PN-A) – Absolute | | | | |
| Change from Baseline to Week 2 | | | | |
| LS Mean <sup>a</sup> | X.XX | x.xx | $x.xxx^b$ | X.XXX <sup>a</sup> |
| LS SD <sup>a</sup> | X.XXX | X.XXX | 711/2/12/12 | x.xxx <sup>c</sup> |
| Median <sup>d</sup> | X.XX | X.XX | | n.n. |
| Min. to Max. <sup>d</sup> | x.x to x.x | x.x to x.x | | |
| Investigator's Global Assessment of Prurigo | | | | |
| Nodularis Activity (IGA PN-A) – Absolute | | | | |
| Change from Baseline to Week 4 | | | | |
| LS Mean <sup>a</sup> | X.XX | X.XX | $x.xxx^b$ | X.XXX <sup>a</sup> |
| LS SD <sup>a</sup> | x.xxx | x.xxx | | x.xxx <sup>c</sup> |
| Median <sup>d</sup> | x.xx | X.XX | | |
| Min. to Max. <sup>d</sup> | x.x to x.x | x.x to x.x | | |
| Investigator's Global Assessment of Prurigo | | | | |
| Nodularis Activity (IGA PN-A) – Absolute | | | | |
| Change from Baseline to Week 10 | | | | |
| LS Mean <sup>a</sup> | x.xx | X.XX | $x.xxx^b$ | x.xxx <sup>a</sup> |
| LS SD <sup>a</sup> | x.xxx | x.xxx | | x.xxx <sup>c</sup> |
| Median <sup>d</sup> | x.xx | X.XX | | |
| Min. to Max. <sup>d</sup> | x.x to x.x | x.x to x.x | | |

<sup>&</sup>lt;sup>a</sup> P-values, least squares means (LS Mean) and standard deviations (LS SD) from an analysis of covariance (ANCOVA) with treatment group and stratification factor as fixed effects, and baseline value as a covariate.

Note: No imputation of missing values. Change calculated as post-baseline – baseline.

<sup>&</sup>lt;sup>b</sup> P-value from a Shapiro-Wilk test for normality.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance (ANCOVA) with treatment group and stratification factor as fixed effects, and baseline value as a covariate.

Table 14.2.3.1: Analysis of Additional Secondary Efficacy Endpoints (Intent-to-Treat Population)


| | Placebo | Serlopitant 5 mg | Normality | Treatment |
|---|---|---|---|---|
| <del>-</del> | (N=xxx) | (N=xxx) | P-Value | P-Value |
| nvestigator's Global Assessment of Prurigo | | | | |
| Nodularis Stage (IGA PN-S) – Absolute Change | | | | |
| rom Baseline to Week 2 | | | _ | |
| LS Mean <sup>a</sup> | X.XX | X.XX | $x.xxx^b$ | x.xxx <sup>a</sup> |
| LS SD <sup>a</sup> | x.xxx | X.XXX | | x.xxx <sup>c</sup> |
| Median <sup>d</sup> | X.XX | X.XX | | |
| Min. to Max. <sup>d</sup> | x.x to x.x | x.x to x.x | | |
| nvestigator's Global Assessment of Prurigo | | | | |
| Nodularis Stage (IGA PN-S) – Absolute Change | | | | |
| rom Baseline to Week 4 | | | | |
| LS Mean <sup>a</sup> | X.XX | X.XX | $x.xxx^b$ | X.XXX <sup>a</sup> |
| LS SD <sup>a</sup> | X.XXX | X.XXX | | x.xxx <sup>c</sup> |
| Median <sup>d</sup> | X.XX | X.XX | | |
| Min. to Max.d | x.x to x.x | x.x to x.x | | |
| nvestigator's Global Assessment of Prurigo | | | | |
| Nodularis Stage (IGA PN-S) – Absolute Change | | | | |
| rom Baseline to Week 10 | | | | |
| LS Mean <sup>a</sup> | X.XX | X.XX | $x.xxx^b$ | x.xxx <sup>a</sup> |
| LS SD <sup>a</sup> | X.XXX | X.XXX | 11111111 | X.XXX <sup>c</sup> |
| Median <sup>d</sup> | X.XX | X.XX | | Α.ΑΑΑ |
| Min. to Max. <sup>d</sup> | x.x to x.x | x.x to x.x | | |

<sup>&</sup>lt;sup>a</sup> P-values, least squares means (LS Mean) and standard deviations (LS SD) from an analysis of covariance (ANCOVA) with treatment group and stratification factor as fixed effects, and baseline value as a covariate.

Note: No imputation of missing values. Change calculated as post-baseline – baseline.

<sup>&</sup>lt;sup>b</sup> P-value from a Shapiro-Wilk test for normality.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance (ANCOVA) with treatment group and stratification factor as fixed effects, and baseline value as a covariate.

Table 14.2.3.1: Analysis of Additional Secondary Efficacy Endpoints (Intent-to-Treat Population)


| | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) | Normality<br>P-Value | Treatment P-Value |
|---|---|---|---|---|
| Dermatology Life Quality Index (DLQI) – | | | | |
| Absolute Change from Baseline to Week 10 | | | | |
| LS Mean <sup>a</sup> | X.XX | X.XX | $x.xxx^b$ | x.xxx <sup>a</sup> |
| LS SD <sup>a</sup> | x.xxx | X.XXX | | x.xxx <sup>c</sup> |
| Median <sup>d</sup> | X.XX | X.XX | | |
| Min. to Max. <sup>d</sup> | x.x to x.x | x.x to x.x | | |
| Dermatology Life Quality Index (DLQI) | | | | |
| Question 1 – Absolute Change from Baseline to | | | | |
| Week 10 | | | | |
| LS Mean <sup>a</sup> | X.XX | X.XX | $\mathbf{x}.\mathbf{x}\mathbf{x}^{\mathbf{b}}$ | x.xxx <sup>a</sup> |
| LS SD <sup>a</sup> | x.xxx | x.xxx | | x.xxx <sup>c</sup> |
| Median <sup>d</sup> | X.XX | X.XX | | |
| Min. to Max.d | x.x to x.x | x.x to x.x | | |

<sup>&</sup>lt;sup>a</sup> P-values, least squares means (LS Mean) and standard deviations (LS SD) from an analysis of covariance (ANCOVA) with treatment group and stratification factor as fixed effects, and baseline value as a covariate.

Note: No imputation of missing values. Change calculated as post-baseline – baseline.

<sup>&</sup>lt;sup>b</sup> P-value from a Shapiro-Wilk test for normality.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance (ANCOVA) with treatment group and stratification factor as fixed effects, and baseline value as a covariate.

Repeat Table 14.2.3.1 for the following:

Table 14.2.3.2: Analysis of Additional Secondary Efficacy Endpoints (Per-Protocol Population)

Table 14.2.4.1: Summary of Worst Itch Numeric Rating Scale (WI-NRS)
(Intent-to-Treat Population)


| WI-NRS | Placebo (N=xxx) | Serlopitant 5 mg (N=xxx) |
|--------------|-----------------|--------------------------|
| Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | x.xx |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics represent average values, obtained by averaging the summary statistics generated from each imputed dataset. Change calculated as post-baseline – baseline.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.4.1: Summary of Worst Itch Numeric Rating Scale (WI-NRS)
(Intent-to-Treat Population)


| NVI NIDO | Placebo | Serlopitant 5 mg |
|---|---|---|
| WI-NRS<br>Week 1 | (N=xxx) | (N=xxx) |
| n | XXX | xxx |
| Mean | X.XX<br>X.XX | XXX<br>X.XX |
| SD | X.XX<br>X.XXX | X.XXX<br>X.XXX |
| Median | | X.XXX<br>X.XX |
| Min. to Max. | x.xx<br>x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | λ.λ ω λ.λ | A.A 10 A.A |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| >= 3 Point Reduction from Baseline | xx.xx% | xx.xx% |
| >= 4 Point Reduction from Baseline | XX.XX% | XX.XX% |
| Week 2 | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | x.xxx |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| >= 3 Point Reduction from Baseline | XX.XX <sup>0</sup> / <sub>0</sub> | XX.XX <sup>0</sup> / <sub>0</sub> |
| >= 4 Point Reduction from Baseline | XX.XX <sup>0</sup> /o | xx.xx% |

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics represent average values, obtained by averaging the summary statistics generated from each imputed dataset. Change calculated as post-baseline – baseline.

Table 14.2.4.1: Summary of Worst Itch Numeric Rating Scale (WI-NRS)
(Intent-to-Treat Population)


| MAL NIDO | Placebo | Serlopitant 5 mg |
|---|---|---|
| WI-NRS<br>Week 3 | (N=xxx) | (N=xxx) |
| | VVV | VVV |
| n<br>Mean | XXX | XXX |
| SD | X.XX | X.XX |
| Median | X.XXX | X.XXX |
| Min. to Max. | X.XX | X.XX |
| | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | XXX | XXX |
| Mean | | |
| SD | X.XX | X.XX |
| Median | X.XXX | X.XXX |
| Min. to Max. | X.XX | X.XX |
| >= 3 Point Reduction from Baseline | x.x to x.x<br>xx.xx% | x.x to x.x<br>xx.xx% |
| >= 4 Point Reduction from Baseline | | |
| | xx.xx% | xx.xx% |
| Week 4 | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| >= 3 Point Reduction from Baseline | xx.xx% | xx.xx% |
| >= 4 Point Reduction from Baseline | XX.XX <sup>0</sup> / <sub>0</sub> | XX.XX <sup>0</sup> / <sub>0</sub> |

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics represent average values, obtained by averaging the summary statistics generated from each imputed dataset. Change calculated as post-baseline – baseline.

Table 14.2.4.1: Summary of Worst Itch Numeric Rating Scale (WI-NRS)
(Intent-to-Treat Population)


| NVI NIDO | Placebo | Serlopitant 5 mg |
|------------------------------------|--------------------|--------------------|
| WI-NRS<br>Week 5 | (N=xxx) | (N=xxx) |
| n | XXX | XXX |
| Mean | X.XX<br>X.XX | XXX<br>X.XX |
| SD | X.XX<br>X.XXX | X.XX<br>X.XXX |
| Median | | X.XXX<br>X.XX |
| Min. to Max. | x.xx<br>x.x to x.x | x.xx<br>x.x to x.x |
| Absolute Change from Baseline | X.X 10 X.X | X.X 10 X.X |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| >= 3 Point Reduction from Baseline | xx.xx% | XX.XX% |
| >= 4 Point Reduction from Baseline | XX.XX% | XX.XX% |
| Week 6 | <b></b> , v | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | x.xx |
| SD | X.XXX | X.XXX |
| Median | X.XX | x.xx |
| Min. to Max. | x.x to x.x | x.x to x.x |
| >= 3 Point Reduction from Baseline | xx.xx% | xx.xx% |
| >= 4 Point Reduction from Baseline | xx.xx% | xx.xx% |

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics represent average values, obtained by averaging the summary statistics generated from each imputed dataset. Change calculated as post-baseline – baseline.

Table 14.2.4.1: Summary of Worst Itch Numeric Rating Scale (WI-NRS)
(Intent-to-Treat Population)


| NVI NIDO | Placebo | Serlopitant 5 mg |
|---|---|---|
| WI-NRS | (N=xxx) | (N=xxx) |
| Week 7 | VVV | VVV |
| n<br>Mean | XXX | XXX |
| SD | X.XX | X.XX |
| Median | X.XXX | X.XXX |
| Min. to Max. | X.XX | X.XX |
| | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline n | XXX | XXX |
| Mean | | |
| SD | X.XX | X.XX |
| Median | X.XXX | X.XXX |
| Min. to Max. | X.XX | X.XX |
| >= 3 Point Reduction from Baseline | x.x to x.x<br>xx.xx% | x.x to x.x<br>xx.xx% |
| >= 4 Point Reduction from Baseline | | |
| | xx.xx% | xx.xx% |
| Week 8 | | |
| n<br>M | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| >= 3 Point Reduction from Baseline | xx.xx% | xx.xx% |
| >= 4 Point Reduction from Baseline | XX.XX <sup>0</sup> / <sub>0</sub> | XX.XX <sup>0</sup> / <sub>0</sub> |

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics represent average values, obtained by averaging the summary statistics generated from each imputed dataset. Change calculated as post-baseline – baseline.

Table 14.2.4.1: Summary of Worst Itch Numeric Rating Scale (WI-NRS)
(Intent-to-Treat Population)


| NVI NIDO | Placebo | Serlopitant 5 mg |
|---|---|---|
| WI-NRS | (N=xxx) | (N=xxx) |
| Week 9 | | |
| n<br>Mari | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| N | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| >= 3 Point Reduction from Baseline | XX.XX <sup>0</sup> / <sub>0</sub> | XX.XX% |
| >= 4 Point Reduction from Baseline | XX.XX <sup>0</sup> ⁄0 | XX.XX% |
| Week 10 | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | x.xxx |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| >= 3 Point Reduction from Baseline | XX.XX <sup>0</sup> /o | xx.xx <sup>0</sup> / <sub>0</sub> |
| >= 4 Point Reduction from Baseline | XX.XX <sup>0</sup> /o | XX.XX <sup>0</sup> / <sub>0</sub> |

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics represent average values, obtained by averaging the summary statistics generated from each imputed dataset. Change calculated as post-baseline – baseline.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.4.1 for the following:

Table 14.2.4.2: Summary of Worst Itch Numeric Rating Scale (WI-NRS) (Per-Protocol Population)

Table 14.2.4.3: Summary of Worst Itch Numeric Rating Scale (WI-NRS) – Observed Data with Follow-up (Intent-to-Treat Population with Observed Week 10 Data)


| WI-NRS | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| | (IN-AXX) | (IN-AXX) |
| Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Week 10 | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| >= 3 Point Reduction from Baseline | xx.xx% | xx.xx% |
| >= 4 Point Reduction from Baseline | XX.XX <sup>0</sup> / <sub>0</sub> | xx.xx% |

Note: No imputation of missing values. Change calculated as post-baseline – baseline.

Table 14.2.4.3: Summary of Worst Itch Numeric Rating Scale (WI-NRS) – Observed Data with Follow-up (Intent-to-Treat Population with Observed Week 10 Data)


| WI-NRS | Placebo (N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| 3-Week Follow-up (Observed Data) | (IV-AAA) | (IN-AAA) |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | x.xxx |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| >= 3 Point Reduction from Baseline | xx.xx% | xx.xx% |
| >= 4 Point Reduction from Baseline | xx.xx% | XX.XX <sup>0</sup> / <sub>0</sub> |
| 5-Week Follow-up (Observed Data) | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| >= 3 Point Reduction from Baseline | xx.xx% | xx.xx% |
| >= 4 Point Reduction from Baseline | xx.xx% | xx.xx% |

Note: No imputation of missing values. Change calculated as post-baseline – baseline.

Table 14.2.5.1.1: Summary of Dermatology Life Quality Index (DLQI)
(Intent-to-Treat Population)


| DLQI | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Week 4 | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.5.1.1: Summary of Dermatology Life Quality Index (DLQI) (Intent-to-Treat Population)


| DLQI | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| Week 10 | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | x.xx | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.5.1.1 for the following:

Table 14.2.5.1.2: Summary of Dermatology Life Quality Index (DLQI) (Per-Protocol Population)

Table 14.2.5.2.1: Summary of Dermatology Life Quality Index (DLQI) Individual Questions (Intent-to-Treat Population)


| DLQI Question 1: Over the last week, how itchy, sore, painful or stinging has your skin been? | Placebo (N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| Baseline | (= : =====) | |
| n | XX | XX |
| Very much | xx ( xx.x%) | xx ( xx.x%) |
| A lot | xx ( xx.x%) | xx ( xx.x%) |
| A little | xx (xx.x%) | xx (xx.x%) |
| Not at all | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | |
| n | XX | XX |
| Very much | xx ( xx.x%) | xx ( xx.x%) |
| A lot | xx (xx.x%) | xx (xx.x%) |
| A little | $xx(x^{0})$ | $xx(x^{0})$ |
| Not at all | xx ( xx.x%) | xx ( xx.x%) |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | x.xxx | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline.

Table 14.2.5.2.1: Summary of Dermatology Life Quality Index (DLQI) – Individual Questions (Intent-to-Treat Population)


| DLQI Question 1: Over the last week, how itchy, sore, painful or stinging has your skin been? Week 10 | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| n | XX | XX |
| Very much | xx ( xx.x%) | xx ( xx.x%) |
| A lot | xx ( xx.x%) | xx ( xx.x%) |
| A little | xx ( xx.x%) | xx (xx.x%) |
| Not at all | xx ( xx.x%) | xx ( xx.x%) |
| n | xxx | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

#### **Include all questions:**

Question 2: Over the last week, how embarrassed or self-conscious have you been because of your skin?

Question 3: Over the last week, how much has your skin interfered with you going shopping or looking after your home or yard?

Question 4: Over the last week, how much has your skin influenced the clothes you wear?

Question 5: Over the last week, how much has your skin affected any social or leisure activities?

Question 6: Over the last week, how much has your skin made it difficult for you to do any sport?

Question 7: Over the last week, has your skin prevented you from working or studying?

Question 8: Over the last week, how much has your skin created problems with your partner or any of your close friends or relatives?

Question 9: Over the last week, how much has your skin caused any sexual difficulties?

Question 10: Over the last week, how much of a problem has the treatment for your skin been, for example by making your home messy, or by taking up time?

Repeat Table 14.2.5.2.1 for the following:

Table 14.2.5.2.2: Summary of Dermatology Life Quality Index (DLQI) – Individual Questions (Per-Protocol Population)

Table 14.2.6.1: Summary of Investigator's Global Assessment of Prurigo Nodularis Activity (IGA PN-A)
(Intent-to-Treat Population)


| | · | |
|-------------------------------|-------------|------------------|
| TG ( 727 ) | Placebo | Serlopitant 5 mg |
| IGA PN-A | (N=xxx) | (N=xxx) |
| Baseline | | |
| N | XX | XX |
| Grade 0 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| Week 2 | | |
| n | XX | XX |
| Grade 0 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx (xx.x%) | xx (xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| n | XXX | xxx |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.6.1: Summary of Investigator's Global Assessment of Prurigo Nodularis Activity (IGA PN-A)
(Intent-to-Treat Population)


| IGA PN-A | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| Week 4 | | |
| n | XX | XX |
| Grade 0 | XX ( XX.X%) | XX ( XX.X%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| n | XXX | xxx |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

Table 14.2.6.1: Summary of Investigator's Global Assessment of Prurigo Nodularis Activity (IGA PN-A)
(Intent-to-Treat Population)


| | Placebo | Serlopitant 5 mg |
|-------------------------------|-------------|------------------|
| IGA PN-A | (N=xxx) | (N=xxx) |
| Week 10 | | |
| n | XX | XX |
| Grade 0 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| n | XXX | xxx |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

Table 14.2.6.1: Summary of Investigator's Global Assessment of Prurigo Nodularis Activity (IGA PN-A)
(Intent-to-Treat Population)


| GA PN-A | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| 3-Week Follow-up | | |
| n | XX | XX |
| Grade 0 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| n | XXX | xxx |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

Table 14.2.6.1: Summary of Investigator's Global Assessment of Prurigo Nodularis Activity (IGA PN-A)
(Intent-to-Treat Population)


| IGA PN-A | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| 5-Week Follow-up | | |
| n | XX | XX |
| Grade 0 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

Table 14.2.6.1: Summary of Investigator's Global Assessment of Prurigo Nodularis Activity (IGA PN-A)

(Intent-to-Treat Population)


| IGA PN-A | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| Latest Follow-up | | |
| n | XX | XX |
| Grade 0 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.6.1 for the following:

Table 14.2.6.2: Summary of Investigator's Global Assessment of Prurigo Nodularis Activity (IGA PN-A) (Per-Protocol Population)

Table 14.2.7.1: Summary of Investigator's Global Assessment of Prurigo Nodularis Stage (IGA PN-S)

(Intent-to-Treat Population)


| IGA PN-S | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| Baseline | (1. 1211) | (1. 11111) |
| n | XX | XX |
| Grade 0 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx (xx.x%) |
| Grade 2 | xx ( xx.x%) | xx (xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| Week 2 | | |
| n | XX | XX |
| Grade 0 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)
Table 14.2.7.1: Summary of Investigator's Global Assessment of Prurigo Nodularis Stage (IGA PN-S)
(Intent-to-Treat Population)


| IGA PN-S | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| Week 4 | | |
| n | XX | XX |
| Grade 0 | XX ( XX.X%) | xx ( xx.x%) |
| Grade 1 | XX ( XX.X%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| n | XXX | xxx |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

Table 14.2.7.1: Summary of Investigator's Global Assessment of Prurigo Nodularis Stage (IGA PN-S)
(Intent-to-Treat Population)


| IGA PN-S | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| Week 10 | | |
| n | XX | XX |
| Grade 0 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| n | XXX | xxx |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

Table 14.2.7.1: Summary of Investigator's Global Assessment of Prurigo Nodularis Stage (IGA PN-S)

(Intent-to-Treat Population)


| IGA PN-S | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| 3-Week Follow-up | | |
| n | XX | XX |
| Grade 0 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

Table 14.2.7.1: Summary of Investigator's Global Assessment of Prurigo Nodularis Stage (IGA PN-S)

(Intent-to-Treat Population)


| GA PN-S | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| -Week Follow-up | | - |
| n | XX | XX |
| Grade 0 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| n | XXX | xxx |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | x.xxx |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

Table 14.2.7.1: Summary of Investigator's Global Assessment of Prurigo Nodularis Stage (IGA PN-S)

(Intent-to-Treat Population)


| IGA PN-S | Placebo<br>(N=xxx) | Serlopitant 5 mg<br>(N=xxx) |
|---|---|---|
| Latest Follow-up | | |
| n | XX | XX |
| Grade 0 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| n | XXX | xxx |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |
| Absolute Change from Baseline | | |
| n | XXX | XXX |
| Mean | X.XX | X.XX |
| SD | X.XXX | X.XXX |
| Median | X.XX | X.XX |
| Min. to Max. | x.x to x.x | x.x to x.x |

Note: No imputation of missing values. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.7.1 for the following:

Table 14.2.7.2: Summary of Investigator's Global Assessment of Prurigo Nodularis Stage (IGA PN-S) (Per-Protocol Population)

Table 14.3.0.1: Summary of Extent of Exposure (Intent-to-Treat Population)

| | Placebo | Serlopitant 5 mg |
|---|---|---|
| | (N=xxx) | N=xxx |
| Total Number of Tablets Useda | • | · |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Total Number of Days of Exposure | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Compliant <sup>b</sup> | | |
| n | XX | XX |
| Yes | xx ( xx.x%) | xx ( xx.x%) |
| No | $xx(x_0^{-1}x$ | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup> Subjects were to dose with 3 tablets on Day 1/Date of First Dose.

Repeat Table 14.3.0.1 for the following:

Table 14.3.0.2: Summary of Extent of Exposure (Per-Protocol Population)

Table 14.3.0.3: Summary of Extent of Exposure (Safety Population)

<sup>&</sup>lt;sup>b</sup> A subject was considered compliant with the dosing regimen if the subject took at least 80% but no more than 120% of expected doses. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.1.1: Overall Summary of Treatment-Emergent Adverse Events (TEAEs) (Safety Population)

| | Placebo | Serlopitant 5 mg |
|---|---|---|
| | (N=xxx) | (N=xxx) |
| Subjects with any TEAE | xx ( xx.x%) | xx ( xx.x%) |
| Number of TEAEs | XX | XX |
| Subjects with any Related TEAE | xx ( xx.x%) | xx ( xx.x%) |
| Number of Related TEAEs | XX | XX |
| Subjects with any Serious TEAE | xx ( xx.x%) | xx ( xx.x%) |
| Number of Serious TEAEs | xx | XX |
| Subjects with any Related Serious TEAE | xx ( xx.x%) | xx ( xx.x%) |
| Number of Related Serious TEAEs | XX | XX |
| Subjects who Died | xx ( xx.x%) | xx ( xx.x%) |
| Subjects who Discontinued Study Drug Due to TEAE | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Severity by Subject | | |
| Grade 5 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Relationship by Subject | | |
| Likely Related | xx ( xx.x%) | xx ( xx.x%) |
| Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) |

Note: TEAEs are AEs with an onset after first dose of study drug.

Table 14.3.1.1.2: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by MedDRA System Organ Class and Preferred Term (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| Total | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class Preferred Term Preferred Term Preferred Term Preferred Term Preferred Term | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

Note: TEAEs are AEs with an onset date after first dose of study drug.

MedDRA Version 21.1.

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more TEAEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Table 14.3.1.1.3: Summary of Treatment-Emergent Adverse Events (TEAEs) Leading to Discontinuation of Study Drug (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | Placebo (N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| Total | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx (xx.x%) | xx ( xx.x%) |
| Preferred Term | xx (xx.x%) | xx ( xx.x%) |
| Preferred Term | xx (xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) |

Note: TEAEs are AEs with an onset date after first dose of study drug.


<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more TEAEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Table 14.3.1.1.4: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population)

| System Organ Class <sup>a</sup> | | Placebo | Serlopitant 5 mg |
|---|---|---|---|
| Preferred Term | Severity <sup>b</sup> | (N=xxx) | (N=xxx) |
| Total | Grade 5 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Grade 5 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Grade 5 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx (xx.x%) |

Note: TEAEs are AEs with an onset after first dose of study drug.


<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more TEAEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

<sup>&</sup>lt;sup>b</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.

Table 14.3.1.1.5: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug
(Safety Population)

| System Organ Class <sup>a</sup><br>Preferred Term | Relationship | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|---|
| Total | Likely Related | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Likely Related | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely Related | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely Related | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more TEAEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.

Note: TEAEs are AEs with an onset after first dose of study drug.


Table 14.3.1.2.1.1: Overall Summary of Post-Drug Adverse Event (AEs) (Safety Population)

| | | Placebo | | | Serlopitant 5 mg | |
|---|---|---|---|---|---|---|
| | Males | Females | Overall | Males | Females | Overall |
| | N=xxx | N=xxx | N=xxx | N=xxx | N=xxx | N=xxx |
| Subjects with any Post-Drug AE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Post-Drug AEs | XX | XX | XX | XX | XX | XX |
| Subjects with any Related Post-Drug AE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Related Post-Drug AEs | XX | XX | XX | XX | XX | XX |
| Subjects with any Serious Post-Drug AE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Serious Post-Drug AEs | xx | XX | XX | XX | xx | xx |
| Subjects with any Related Serious Post-Drug AE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Related Serious Post-Drug AEs | xx | xx | xx | XX | xx | xx |
| Subjects who Died | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Severity by Subject | | | | | | |
| Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Relationship by Subject | | | | | | |
| Likely Related | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Table includes AEs with an onset after last dose of study drug.

Table 14.3.1.2.1.2: Overall Summary of Post-Drug Adverse Events (AEs) Occurring 1-7 Days Post Last Dose (Safety Population)

| | Placebo | Serlopitant 5 mg |
|---|---|---|
| | (N=xxx) | (N=xxx) |
| Subjects with any Post-Drug AE | xx ( xx.x%) | xx ( xx.x%) |
| Number of Post-Drug AEs | XX | XX |
| Subjects with any Related Post-Drug AE | xx ( xx.x%) | xx ( xx.x%) |
| Number of Related Post-Drug AEs | XX | xx |
| Subjects with any Serious Post-Drug AE | xx ( xx.x%) | xx ( xx.x%) |
| Number of Serious Post-Drug AEs | XX | xx |
| Subjects with any Related Serious Post-Drug AE | xx ( xx.x%) | xx ( xx.x%) |
| Number of Related Serious Post-Drug AEs | XX | XX |
| Subjects who Died | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Severity by Subject | | |
| Grade 5 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Relationship by Subject | | |
| Likely Related | xx ( xx.x%) | xx ( xx.x%) |
| Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) |

Note: Table includes AEs with an onset date within 1 to 7 days after last dose of study drug. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.3.1.2.1.2 for the following, with adjusted foonotes:

Table 14.3.1.2.1.3: Overall Summary of Post-Drug Adverse Events (AEs) Occurring 8-14 Days Post Last Dose (Safety Population)

Note: Table includes AEs with an onset date within 8 to 14 days after last dose of study drug.

Table 14.3.1.2.1.4: Overall Summary of Post-Drug Adverse Events (AEs) Occurring 15-21 Days Post Last Dose (Safety Population)

Note: Table includes AEs with an onset date within 15 to 21 days after last dose of study drug.

Table 14.3.1.2.1.5: Overall Summary of Post-Drug Adverse Events (AEs) Occurring 22-28 Days Post Last Dose (Safety Population)

Note: Table includes AEs with an onset date within 22 to 28 days after last dose of study drug.

Table 14.3.1.2.1.6: Overall Summary of Post-Drug Adverse Events (AEs) Occurring 29-35 Days Post Last Dose (Safety Population)

Note: Table includes AEs with an onset date within 29 to 35 days after last dose of study drug.

Table 14.3.1.2.2.1: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) by MedDRA System Organ Class and Preferred Term (Safety Population)


| | | Placebo | | | Serlopitant 5 mg | |
|---|---|---|---|---|---|---|
| System Organ Class <sup>a</sup> Preferred Term | Males<br>(N=xxx) | Females (N=xxx) | Overall (N=xxx) | Males<br>(N=xxx) | Females (N=xxx) | Overall (N=xxx) |
| Total | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class Preferred Term Preferred Term Preferred Term Preferred Term | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more AEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Note: Table includes AEs with an onset after last dose of study drug.


Table 14.3.1.2.2: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 1-7 Days Post Last Dose by MedDRA System Organ Class and Preferred Term

(Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| Total | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class Preferred Term Preferred Term Preferred Term Preferred Term | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more AEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Note: Table includes AEs with an onset date within 1 to 7 days after last dose of study drug.


Repeat Table 14.3.1.2.2.2 for the following, with adjusted foonotes:

Table 14.3.1.2.2.3: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 8-14 Days Post Last Dose by MedDRA System Organ Class and Preferred Term (Safety Population)

Note: Table includes AEs with an onset date within 8 to 14 days after last dose of study drug.

Table 14.3.1.2.2.4: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 15-21 Days Post Last Dose by MedDRA System Organ Class and Preferred Term (Safety Population)

Note: Table includes AEs with an onset date within 15 to 21 days after last dose of study drug.

Table 14.3.1.2.2.5: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 22-28 Days Post Last Dose by MedDRA System Organ Class and Preferred Term (Safety Population)

Note: Table includes AEs with an onset date within 22 to 28 days after last dose of study drug.

Table 14.3.1.2.2.6: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 29-35 Days Post Last Dose by MedDRA System Organ Class and Preferred Term (Safety Population)

Note: Table includes AEs with an onset date within 29 to 35 days after last dose of study drug.

Table 14.3.1.2.3.1: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) by Severity (Safety Population)

| | | | Placebo | | | Serlopitant 5 mg | |
|---|---|---|---|---|---|---|---|
| System Organ Class <sup>a</sup> | | Males | Females | Overall | Males | Females | Overall |
| Preferred Term | Severity <sup>b</sup> | (N=xxx) | N=xxx | N=xxx | (N=xxx) | N=xxx | N=xxx |
| Total | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more AEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

Note: Table includes AEs with an onset after last dose of study drug.


<sup>&</sup>lt;sup>b</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.

Table 14.3.1.2.3.2: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 1-7 Days Post Last Dose by Severity (Safety Population)


| System Organ Class <sup>a</sup> | | Placebo | Serlopitant 5 mg |
|---|---|---|---|
| Preferred Term | Severity <sup>b</sup> | (N=xxx) | (N=xxx) |
| Total | Grade 5 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Grade 5 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Grade 5 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx (xx.x%) |

Note: Table includes AEs with an onset date within 1 to 7 days after last dose of study drug.


<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more AEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

<sup>&</sup>lt;sup>b</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.

Repeat Table 14.3.1.2.3.2 for the following, with adjusted foonotes:

Table 14.3.1.2.3.3: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 8-14 Days Post Last Dose by Severity (Safety Population)

Note: Table includes AEs with an onset date within 8 to 14 days after last dose of study drug.

Table 14.3.1.2.3.4: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 15-21 Days Post Last Dose by Severity (Safety Population)

Note: Table includes AEs with an onset date within 15 to 21 days after last dose of study drug.

Table 14.3.1.2.3.5: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 22-28 Days Post Last Dose by Severity (Safety Population)

Note: Table includes AEs with an onset date within 22 to 28 days after last dose of study drug.

Table 14.3.1.2.3.6: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 29-35 Days Post Last Dose by Severity (Safety Population)

Note: Table includes AEs with an onset date within 29 to 35 days after last dose of study drug.

Table 14.3.1.2.4.1: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) by Relationship to Study Drug (Safety Population) (Page 1 of xx)

| | | | Placebo | | | Serlopitant 5 mg | |
|---|---|---|---|---|---|---|---|
| System Organ Class <sup>a</sup> | D 1 2 12 | Males | Females | Overall | Males | Females | Overall |
| Preferred Term | Relationship | (N=xxx) | N=xxx | (N=xxx) | N=xxx | (N=xxx) | N=xxx |
| Total | Likely Related | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Likely Related | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely Related | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely Related | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more AEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.

Note: Table includes AEs with an onset after last dose of study drug.


Table 14.3.1.2.4.2: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 1-7 Days Post Last Dose by Relationship to Study Drug (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | Relationship | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|---|
| Total | Likely Related | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Likely Related | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely Related | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely Related | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more AEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.

Note: Table includes AEs with an onset date within 1 to 7 days after last dose of study drug. MedDRA Version 21.1.

Repeat Table 14.3.1.2.4.2 for the following, with adjusted foonotes:

Table 14.3.1.2.4.3: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 8-14 Days Post Last Dose by Relationship to Study Drug (Safety Population)

Note: Table includes AEs with an onset date within 8 to 14 days after last dose of study drug.

Table 14.3.1.2.4.4: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 15-21 Days Post Last Dose by Relationship to Study Drug (Safety Population)

Note: Table includes AEs with an onset date within 15 to 21 days after last dose of study drug.

Table 14.3.1.2.4.5: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 22-28 Days Post Last Dose by Relationship to Study Drug (Safety Population)

Note: Table includes AEs with an onset date within 22 to 28 days after last dose of study drug.

Table 14.3.1.2.4.6: Summary of Subjects Reporting Post-Drug Adverse Events (AEs) Occurring 29-35 Days Post Last Dose by Relationship to Study Drug (Safety Population)

Note: Table includes AEs with an onset date within 29 to 35 days after last dose of study drug.

Table 14.3.1.3.1: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by MedDRA System Organ Class and Preferred Term (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| Total | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class Preferred Term Preferred Term Preferred Term Preferred Term Preferred Term | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

Note: TEAEs are AEs with an onset date after first dose of study drug.


<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more TEAEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Table 14.3.1.3.2: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population)


| System Organ Class <sup>a</sup> | | Placebo | Serlopitant 5 mg |
|---|---|---|---|
| Preferred Term | <u>Severity</u> | (N=xxx) | (N=xxx) |
| Total | Grade 5 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Grade 5 | xx ( xx.x%) | xx ( xx.x%) |
| , | Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx (xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Grade 5 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) |

Note: TEAEs are AEs with an onset after first dose of study drug.


<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more serious TEAEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

<sup>&</sup>lt;sup>b</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.

Table 14.3.1.3.3: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | Relationship | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|---|
| Total | Likely Related | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Likely Related | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely Related | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely Related | xx ( xx.x%) | xx ( xx.x%) |
| | Likely Unrelated | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more TEAEs that map to the MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.

Note: TEAEs are AEs with an onset after first dose of study drug.


Table 14.3.1.4.1.1: Summary of Hematology Laboratory Results (Safety Population)

| | Placebo | Serlopitant 5 mg |
|-----------------------------------------|----------|------------------|
| | (N=xxx) | (N=xxx) |
| <test name=""> (<units>)</units></test> | | |
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Absolute Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Note: No imputation of missing values. Baseline is the latest recorded value prior to first dose of study drug. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table to include post-baseline visits of "Week 2", "Week 10", "3-Week Follow-up", "5-Week Follow-up", "Latest Follow-up".

Table to include following lab tests: "BASOPHILS", "EOSINOPHILS", "HCT", "HGB", "LYMPHOCYTES", "MCH", "MCHC", "MCV", "MONOCYTES", "NEUTROPHILS", "PLATELET COUNT", "RBC", "WBC".

Table 14.3.1.4.1.2: Shift Summary of Hematology Laboratory Results (Safety Population)

| <test name=""> (<units>)</units></test> | | Placebo<br>(N=xxx) | | | Serlopitant 5 mg<br>(N=xxx) | |
|---|---|---|---|---|---|---|
| | | Week 2 | | | Week 2 | |
| Baseline | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Week 10 | | | | Week 10 | |
| Baseline | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | 3- | 3-Week Follow-up | | | 3-Week Follow-up | |
| <u>Baseline</u> | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | -Week Follow-up | | 5-Week Follow-up | | |
| <u>Baseline</u> | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Latest Follow-up | | | | atest Follow-up | |
| <u>Baseline</u> | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: BNL=Below Normal Limit, WNL=Within Normal Limits, ANL=Above Normal Limit.

No imputation of missing values. Baseline is the latest recorded value prior to first dose of study drug. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table to include the same lab tests used in Table 14.3.1.4.1.1.

Table 14.3.1.4.2.1: Summary of Chemistry Laboratory Results (Safety Population)

| | DI 1 | 0.1.1.1. |
|-----------------------------------------|----------|------------------|
| | Placebo | Serlopitant 5 mg |
| | (N=xxx) | (N=xxx) |
| <test name=""> (<units>)</units></test> | | |
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Absolute Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Note: No imputation of missing values. Baseline is the latest recorded value prior to first dose of study drug. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table to include post-baseline visits of "Week 2", "Week 10", "3-Week Follow-up", "5-Week Follow-up", "Latest Follow-up".

Table to include following lab tests: "ALBUMIN", "ALKALINE PHOSPHATASE", "ALT", "AST", "BICARBONATE", "BILIRUBIN, TOTAL", "BUN", "CALCIUM", "CHLORIDE", "CHOLESTEROL, TOTAL", "CREATININE", "GLUCOSE, RANDOM", "HDL-CHOLESTEROL", "LDH", "LDL-CHOLESTEROL", "MAGNESIUM", "PHOSPHORUS", "POTASSIUM", "PROTEIN, TOTAL", "SODIUM", "TRIGLYCERIDES", "URIC ACID".

Table 14.3.1.4.2.2: Shift Summary of Chemistry Laboratory Results (Safety Population)

| <test name=""> (<units>)</units></test> | | Placebo<br>(N=xxx) | | | Serlopitant 5 mg<br>(N=xxx) | |
|---|---|---|---|---|---|---|
| | | Week 2 | | | Week 2 | |
| Baseline | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | Week 10 | | | Week 10 | |
| Baseline | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | 3- | Week Follow-up | | 3. | -Week Follow-up | |
| Baseline | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | 5- | Week Follow-up | | 5 | -Week Follow-up | |
| <u>Baseline</u> | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | I | atest Follow-up | | I | Latest Follow-up | |
| <u>Baseline</u> | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: BNL=Below Normal Limit, WNL=Within Normal Limits, ANL=Above Normal Limit.

No imputation of missing values. Baseline is the latest recorded value prior to first dose of study drug. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table to include the same lab tests used in Table 14.3.1.4.2.1.

Table 14.3.1.4.3.1.1: Summary of Endocrine/Reproductive Endocrine Laboratory Results (Safety Population)

| | Placebo | Serlopitant 5 mg |
|-----------------------------------------|----------|------------------|
| | (N=xxx) | (N=xxx) |
| <test name=""> (<units>)</units></test> | | · · |
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 10 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Absolute Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Note: No imputation of missing values. Baseline is the latest recorded value prior to first dose of study drug. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table to include post-baseline visits of "Week 10", "3-Week Follow-up", "5-Week Follow-up", "Latest Follow-up".

Table to include following lab tests: "TSH ULTRASENSITIVE", "THYROXINE, FREE", "CORTISOL, SERUM RANDOM", "ACTH, PLASMA", "ANTI-MULLERIAN HORMONE", "FSH", "ESTRADIOL", "LUTEINIZING HORMONE", "PROGESTERONE".

Table 14.3.1.4.3.1.2: Summary of Reproductive Endocrine Laboratory Results (Safety Population – Females Using Hormonal Contraception/Therapy) (Page 1 of xx)

| | Placebo | Serlopitant 5 mg |
|-----------------------------------------|----------|------------------|
| | (N=xxx) | (N=xxx) |
| <test name=""> (<units>)</units></test> | | |
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 10 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Absolute Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Note: No imputation of missing values. Baseline is the latest recorded value prior to first dose of study drug. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table to include post-baseline visits of "Week 10", "3-Week Follow-up", "5-Week Follow-up", "Latest Follow-up".

Table to include following lab tests: "ANTI-MULLERIAN HORMONE", "FSH", "ESTRADIOL", "LUTEINIZING HORMONE", "PROGESTERONE".

Table 14.3.1.4.3.1.3: Summary of Reproductive Endocrine Laboratory Results (Safety Population – Females Not Using Hormonal Contraception/Therapy) (Page 1 of xx)

| | Placebo | Serlopitant 5 mg |
|-----------------------------------------|----------|------------------|
| | (N=xxx) | (N=xxx) |
| <test name=""> (<units>)</units></test> | | |
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 10 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Absolute Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Note: No imputation of missing values. Baseline is the latest recorded value prior to first dose of study drug. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table to include post-baseline visits of "Week 10", "3-Week Follow-up", "5-Week Follow-up", "Latest Follow-up".

Table to include following lab tests: "ANTI-MULLERIAN HORMONE", "FSH", "ESTRADIOL", "LUTEINIZING HORMONE", "PROGESTERONE".

Table 14.3.1.4.3.2: Shift Summary of Endocrine/Reproductive Endocrine Laboratory Results
(Safety Population)

| <test name=""> (<units>)</units></test> | | Placebo<br>(N=xxx) | | | Serlopitant 5 mg<br>(N=xxx) | |
|---|---|---|---|---|---|---|
| | | Week 10 | | | Week 10 | |
| Baseline | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | 3- | -Week Follow-up | | 3- | -Week Follow-up | |
| Baseline | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | 5 | -Week Follow-up | | 5- | -Week Follow-up | |
| <u>Baseline</u> | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | I | Latest Follow-up | | I | Latest Follow-up | |
| <u>Baseline</u> | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: BNL=Below Normal Limit, WNL=Within Normal Limits, ANL=Above Normal Limit.

No imputation of missing values. Baseline is the latest recorded value prior to first dose of study drug. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table to include following lab tests: "TSH ULTRASENSITIVE", "THYROXINE, FREE", "CORTISOL, SERUM RANDOM", "ACTH, PLASMA", "ANTI-MULLERIAN HORMONE".

Table 14.3.1.5.1.1: Summary of Treatment-Emergent Electrocardiogram (ECG) Parameter Abnormalities (Safety Population)


| | Placebo | Serlopitant 5 mg |
|---|---|---|
| | (N=xxx) | (N=xxx) |
| Number of Subjects with Treatment-Emergent ECG Results | XXX | XXX |
| PR Interval | | |
| > 200 msec | xx (xx.x%) | xx ( xx.x%) |
| > 220 msec | xx ( xx.x%) | xx ( xx.x%) |
| Change from Baseline in PR Interval | | |
| >= 25% and $> 200$ msec | xx ( xx.x%) | xx ( xx.x%) |
| QRS Interval | | |
| > 110 msec | xx (xx.x%) | xx (xx.x%) |
| > 120 msec | xx ( xx.x%) | xx ( xx.x%) |
| Change from Baseline in QRS Interval | | |
| >= 25% and $> 110$ msec | xx (xx.x%) | xx ( xx.x%) |
| >= 25% and $> 120$ msec | xx ( xx.x%) | xx ( xx.x%) |
| QTcF Interval | | |
| > 450 - 470 msec | xx (xx.x%) | xx (xx.x%) |
| > 470 - 500 msec | xx ( xx.x%) | xx ( xx.x%) |
| > 500 msec | xx ( xx.x%) | xx ( xx.x%) |
| Change from Baseline in QTcF Interval | | |
| > 30 - 60 msec | xx (xx.x%) | xx ( xx.x%) |
| > 60 msec | xx ( xx.x%) | xx ( xx.x%) |
| QTcF Interval > 500 msec and Change from Baseline > 60 msec | xx ( xx.x%) | xx ( xx.x%) |

Note: No imputation of missing values. Baseline is the latest recorded value prior to first dose of study drug. Change calculated as post-baseline – baseline. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.5.1.1: Summary of Treatment-Emergent Electrocardiogram (ECG) Abnormalities (Safety Population)


| Number of Subjects with Treetment Emergent ECG | Placebo<br>(N=xxx) | Serlopitant 5 mg (N=xxx) |
|---|---|---|
| Number of Subjects with Treatment-Emergent ECG<br>Results | XXX | XXX |
| QTcB Interval | | |
| > 450 - 470 msec | xx ( xx.x%) | xx ( xx.x%) |
| > 470 - 500 msec | xx ( xx.x%) | xx (xx.x%) |
| > 500 msec | xx ( xx.x%) | xx ( xx.x%) |
| Change from Baseline in QTcB Interval | | |
| > 30 - 60 msec | xx ( xx.x%) | xx ( xx.x%) |
| > 60 msec | xx ( xx.x%) | xx ( xx.x%) |
| QTcB Interval > 500 msec and Change from Baseline > 60 msec | xx ( xx.x%) | xx ( xx.x%) |

Note: No imputation of missing values. Baseline is the latest recorded value prior to first dose of study drug. Change calculated as post-baseline – baseline. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)
Table 14.3.1.5.1.2: Summary of Electrocardiogram Parameters (Safety Population)

| | Placebo | Serlopitant 5 mg |
|-------------------------------------------|----------|------------------|
| | (N=xxx) | (N=xxx) |
| <parameter> (<units>)</units></parameter> | | |
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Absolute Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Note: No imputation of missing values. Baseline is the latest recorded value prior to first dose of study drug. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table to include parameters "ECG Mean Heart Rate (beats/min)", "PR Interval, Aggregate (msec)", "QRS Duration, Aggregate (msec)", "QT Interval, Aggregate (msec)", "QTcB Interval, Aggregate (msec)", "RR Interval, Aggregate (msec)".

Table to include post-baseline visits of "Week 2", "Week 4", "Week 10", "3-Week Follow-up", "5-Week Follow-up", "Latest Follow-up".

Table 14.3.1.5.1.3: Shift Summary of Overall Electrocardiogram (ECG) Assessments (Safety Population)


| Overall ECG Assessment (per Investigator) | 9 / | | | Serlopitant 5 mg (N=xxx) | | |
|---|---|---|---|---|---|---|
| - ·· | | Week 2 | .1 1 22 | | Week 2 | |
| <u>Baseline</u> | Normal | Abnormal, NCS | Abnormal, CS | Normal | Abnormal, NCS | Abnormal, CS |
| Normal | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Abnormal, NCS | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Abnormal, CS | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | Week 4 | | | Week 4 | |
| <u>Baseline</u> | Normal | Abnormal, NCS | Abnormal, CS | Normal | Abnormal, NCS | Abnormal, CS |
| Normal | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Abnormal, NCS | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Abnormal, CS | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | Week 10 | | | Week 10 | |
| <u>Baseline</u> | Normal | Abnormal, NCS | Abnormal, CS | Normal | Abnormal, NCS | Abnormal, CS |
| Normal | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Abnormal, NCS | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Abnormal, CS | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | 3 | -Week Follow-up | | 3 | -Week Follow-up | |
| <u>Baseline</u> | Normal | Abnormal, NCS | Abnormal, CS | Normal | Abnormal, NCS | Abnormal, CS |
| Normal | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Abnormal, NCS | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Abnormal, CS | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | 5 | -Week Follow-up | | 5 | -Week Follow-up | |
| <u>Baseline</u> | Normal | Abnormal, NCS | Abnormal, CS | Normal | Abnormal, NCS | Abnormal, CS |
| Normal | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Abnormal, NCS | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Abnormal, CS | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: No imputation of missing values. Baseline is the latest recorded value prior to first dose of study drug. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week Follow-up visits.

NCS=Not Clinically Significant; CS=Clinically Significant.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

# Table 14.3.1.5.1.3: Shift Summary of Overall Electrocardiogram (ECG) Assessments (Safety Population) 

| Overall ECG Assessment (per Investigator) | Placebo (N=xxx) Latest Follow-up | | | | Serlopitant 5 mg<br>(N=xxx)<br>Latest Follow-up | |
|---|---|---|---|---|---|---|
| <u>Baseline</u><br>Normal<br>Abnormal, NCS<br>Abnormal, CS | Normal<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | Abnormal, NCS xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) | Abnormal, CS xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) | Normal<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | Abnormal, NCS xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) | Abnormal, CS xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) |

Note: No imputation of missing values. Baseline is the latest recorded value prior to first dose of study drug. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

NCS=Not Clinically Significant; CS=Clinically Significant.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.6.1: Summary of Vital Signs (Safety Population)

| | Placebo | Serlopitant 5 mg |
|-------------------------------------------|----------|------------------|
| | (N=xxx) | (N=xxx) |
| <parameter> (<units>)</units></parameter> | | |
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Absolute Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Note: Baseline is the latest recorded value prior to first dose of study drug. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table to include parameters in following order: "Temperature (degrees Celsius)", "Respiration Rate (breaths/min)", "Heart Rate (beats/min)", "Systolic Blood Pressure (mmHg)", "Diastolic Blood Pressure (mmHg)".

Table to include post-baseline visits of "Week 2", "Week 4", "Week 6", "Week 10", "3-Week Follow-up", "5-Week Follow-up", "Latest Follow-up".

Table 14.3.1.7.1: Summary of Hospital Anxiety and Depression Scale (HADS)

(Safety Population)


| | Placebo | Serlopitant 5 mg |
|-------------------------------|----------|------------------|
| | (N=xxx) | N=xxx |
| Subscale> | | |
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Veek 4 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Absolute Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Note: Baseline is the latest recorded value prior to first dose of study drug. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table to include subscales in following order: "Anxiety Subscale", "Depression Subscale".

Table to include post-baseline visits of "Week 4", "Week 10", "3-Week Follow-up", "5-Week Follow-up", "Latest Follow-up".

Table 14.3.1.8.1: Summary of Epworth Sleepiness Scale (ESS)
(Safety Population)

| | Placebo | Serlopitant 5 mg |
|-------------------------------|----------|------------------|
| | (N=xxx) | (N=xxx) |
| CSS | | |
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Veek 4 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Absolute Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Note: Baseline is the latest recorded value prior to first dose of study drug. Change calculated as post-baseline – baseline. "Latest Follow-up" visit includes the latest available follow-up information for each subject from the 3-Week or 5-Week Follow-up visits.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table to include post-baseline visits of "Week 4", "Week 10", "3-Week Follow-up", "5-Week Follow-up", "Latest Follow-up".

Table 14.3.1.9: Summary of Pharmacokinetic Concentrations (Safety Population)

| | Placebo | Serlopitant 5 mg |
|---------------------------------------|----------|------------------|
| | (N=xxx) | N=xxx |
| <analyte> (<units>)</units></analyte> | , , | , , |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 4 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 10 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Note: No imputation of missing values.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table to include analytes in following order: "M1/M1a", "M2/M2a", "M3", "Serlopitant".

Table 14.3.1.10: Summary of Menstrual Cycles (Safety Population)

| | Placebo | Serlopitant 5 mg |
|------------------------------|----------|------------------|
| | (N=xxx) | (N=xxx) |
| Number of Menstrual Cycles | , | , |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Duration of Menstrual Cycles | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Note: No imputation of missing values.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

## 11. INDEX OF PLANNED LISTINGS

| Listing 16.1.7: Randomization Scheme | 118 |
|---|---|
| Listing 16.2.1.1: Subject Disposition Information | 119 |
| Listing 16.2.1.2: Discontinued Subjects | 120 |
| Listing 16.2.2.1: Inclusion/Exclusion Criteria Not Met | 121 |
| Listing 16.2.3: Analysis Populations | 122 |
| Listing 16.2.4.1: Subject Demographic Information | 123 |
| Listing 16.2.4.2.1: Unique Medical History Coded to MedDRA System Organ Classes and Preferred Terms | 124 |
| Listing 16.2.4.2.2: Medical History | 125 |
| Listing 16.2.4.3.1: Prurigo Nodularis History | 126 |
| Listing 16.2.4.3.2: Prior Therapies | 127 |
| Listing 16.2.4.4.1: Unique Medication Names Coded to WHO DDE ATC Level 2 Terms and Preferred Names | |
| Listing 16.2.4.4.2: Concomitant Medications | 129 |
| Listing 16.2.4.5: Concomitant Procedures/Therapies | 130 |
| Listing 16.2.4.6: Physical Examination | 131 |
| Listing 16.2.5.1: Study Visit/Phone Call Compliance | 132 |
| Listing 16.2.5.2: Study Drug Dispensing and Return | 133 |
| Listing 16.2.5.3: Dosing Deviations | 134 |
| Listing 16.2.6.1.1: Worst Itch Numeric Rating Scale (WI-NRS) at Screening | 135 |
| Listing 16.2.6.1.2: Worst Itch Numeric Rating Scale (WI-NRS) | 136 |
| Listing 16.2.6.2: IGA PN-A and IGA PN-S Results | 137 |
| Listing 16.2.6.3: Dermatology Life Quality Index (DLQI) | 138 |
| Listing 16.2.6.4: Photography | 139 |
| Listing 16.2.7.1.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms | 140 |
| Listing 16.2.7.1.2: Treatment-Emergent Adverse Events | 141 |
| Listing 16.2.7.1.3: Serious Adverse Events | 142 |
| Listing 16.2.7.1.4: Subjects Who Permanently Discontinued Study Drug Due to Adverse Events | 143 |
| Listing 16.2.7.2.1: Hospital Anxiety and Depression Scale | 144 |
| Listing 16.2.7.2.2: Epworth Sleepiness Scale | 145 |

| Listing 16.2.7.3: Menstrual Diary | .146 |
|---|---|
| Listing 16.2.8.1: Pregnancy Test Results. | .147 |
| Listing 16.2.8.2.1: Laboratory Test Results | .148 |
| Listing 16.2.8.2.2: Out of Range Laboratory Results | .149 |
| Listing 16.2.8.2.3: Common Laboratory Comments Including Reference Ranges for Specific Laboratory Tests | |
| Listing 16.2.8.3: Electrocardiogram Test Results | .151 |
| Listing 16.2.8.4: Vital Signs | .152 |
| Listing 16.2.8.5: Pharmacokinetics Blood Sample Collection and Plasma Concentrations | .153 |

## Listing 16.1.7: Randomization Scheme (Page xx of yy)

| Subject | Age/Sex | Evaluable | Randomization<br>Strata | Randomization<br>Date | Assigned<br>Treatment Group | Was the subject previously a Screen Fail? | Previous Screening<br>Subject Number |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxx | xxxxxxxx | ***** | xxx | xxxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxx | xxxxxxxxx | xxxxxx xxxxxx | xxx | xxxxx |
| xxxxxx | XXXX | xxxxxxxx | xxxx | xxxxxxxxx | xxxxxx xxxxxx | xxx | xxxxxx |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject.

Listing 16.2.1.1: Subject Disposition Information
Treatment Group
(Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Evaluable | F: Date of First Dose L: Date of Last Dose | R: Reason for Treatment Discontinuation P: Primary AE Number/Specify | E: Follow-up Discontinuation Date (Day) R: Reason for Follow-up Discontinuation | D: Date of Last Contact P: Primary AE Number/Specify C: Continuing into MTI-107? |
|---|---|---|---|---|
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxx-xx-xx<br>L: xxxx-xx | R: xxxxxxxxx xx xxxxxxxxxxxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) R: xxxxxxxxxx xx xxxxxxxxx | D: xxxx-xx-xx P: xxxxxxxxxx C: xxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxx-xx-xx<br>L: xxxx-xx-xx | R: xxxxxxxxx xx xxxxxxxxxxxxxxxxxxxxxxx | E: xxxx-xx-xx (xx)<br>R: xxxxxxxxx xx xxxxxxxxx | D: xxxx-xx-xx P: xxxxxxxxxx C: xxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxx-xx-xx<br>L: xxxx-xx-xx | R: xxxxxxxx xxxx xxxxxxx xxxxx<br>P: xxxxxxxxxx | E: xxxx-xx-xx (xx) R: xxxx xx xxxxxxxx | D:<br>P: xxxxxxxxxx<br>C: xxx |

## Listing sorted by Subject.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
 date - date of first dose + 1 for dates on or after first dose.
Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

## Listing 16.2.1.2: Discontinued Subjects Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Evaluable | F: Date of First Dose L: Date of Last Dose | R: Reason for Treatment Discontinuation P: Primary AE Number/Specify | E: Follow-up Discontinuation Date (Day)¹ R: Reason for Follow-up Discontinuation | D: Date of Last Contact P: Primary AE Number/Specify C: Continuing into MTI-107? |
|---|---|---|---|---|
| S: xxxxxx | F: xxxx-xx-xx | R: xxxxxxxxx xx xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | D: xxxx-xx-xx |
| A: xxxx<br>E: xxxxxxxxx | L: xxxx-xx-xx | P: xxxxxxxxx | R: xxxxxxxxx xx xxxxxxxxx | P: xxxxxxxxxx<br>C: xxx |
| S: xxxxxx | F: xxxx-xx-xx | R: xxxxxxxxx xx xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | D: xxxx-xx-xx |
| A: xxxx<br>E: xxxxxxxx | L: xxxx-xx-xx | P: xxxxxxxxxx | R: xxxxxxxxx xx xxxxxxxxx | P: xxxxxxxxxx<br>C: xxx |
| S: xxxxxx | F: xxxx-xx-xx | R: xxxxxxxx xxxx xxxxxxx xxxxx | E: xxxx-xx-xx (xx) | D: |
| A: xxxx<br>E: xxxxxxxx | L: xxxx-xx-xx | P: xxxxxxxxx | R: xxxx xx xxxxxxxx | P: xxxxxxxxxx<br>C: xxx |

## Listing sorted by Subject.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
 date - date of first dose + 1 for dates on or after first dose.
Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.2.1: Inclusion/Exclusion Criteria Not Met
Treatment Group
(Page xx of yy)

| Subject | Age/Sex | Evaluable | Criterion Failed | Description |
|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxx | xxxxx xxx xx xxxxxxx xxxx xxxx xxxxxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxx | ***** *** ** ******* **** ************ |
| xxxxxx | xxxx | xxxxxxxx | xxxxx | ***** *** ** ****** *** ************ |
| | | | xxxxx | ***** *** ** ****** *** ************ |
| | | | xxxxx | xxxxx xxx xx xxxxxxxx xxxx xxxx xxxxxxx |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject and Criterion Failed.

## Listing 16.2.3: Analysis Populations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Population | Included | Reason(s) Excluded | Exception(s) |
|---|---|---|---|---|---|
| xxxxxx | xxxx | Intent-to-Treat | XXX | | |
| | | Safety | XXX | | |
| | | Per-Protocol | XX | xxxxxxxxxx xxxxxx xxxxxxxx | |
| xxxxx | xxxx | Intent-to-Treat | XXX | | |
| | | Safety | XXX | | |
| | | Per-Protocol | XXX | | |
| xxxxx | xxxx | Intent-to-Treat | xxx | | |
| | | Safety | XXX | | |
| | | Per-Protocol | XX | xxxxxxxxx xxxxxx xxxxxxx | xxxxxxxxx xxxxxx xxxxxxx |
| | | | | xxxxxxxxx xxxxxxx xxxxxxx | |
| xxxxx | xxxx | Intent-to-Treat | xxx | | |
| | | Safety | XX | xxxxxxxxx xxxxxx xxxxxxx | |
| | | Per-Protocol | XX | xxxxxxxxx xxxxxx xxxxxxx | |
| | | | | XXXXXXXXXX XXXXXXX XXXXXXXX | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject and Population (as ordered above).

Listing 16.2.4.1: Subject Demographic Information
Treatment Group
(Page xx of yy)

| Subject | Evaluable | B: Date of E<br>A: Age<br>S: Sex | Birth<br>R: Race<br>E: Ethnicity | C: Childbearing Potential M: Method of Contraceptio | <pre>I: Informed Consent Date/Protocol Version n P: Did subject consent to photography?</pre> |
|---|---|---|---|---|---|
| xxxxxx | xxxxxxxx | B: xxxx-xx-x<br>A: xx<br>S: xxxxxx | R: xxxxxx xxxxxxxx<br>xx xxxxx xxxxxxx<br>xxxxxx | C: xxx M: xxxxxxxxxx xxxxxxxx xxxxxxxxxx | I: V2.1/xxxx-xx-xx<br>V3/xxxx-xx-xx<br>x P: xxx |
| xxxxxx | xxxxxxxx | B: xxxx-xx-x<br>A: xx<br>S: xxxx | R: XXXXX<br>E: XXXXXXXX XX XXXXX | C: xx<br>M: | I: V2/xxxx-xx-xx<br>P: xxx |
| xxxxx | xxxxxxxx | B: xxxx-xx-x<br>A: xx<br>S: xxxxx | R: XXXXX<br>E: XXXXXXXX XX XXXXX | C: xxx<br>M: xxxxxxxx xxxxxxxxxxxx | I: V3/xxxx-xx-xx<br>P: xxx |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject. Include all instances of informed consents and associated protocol versions.

Listing 16.2.4.2.1: Unique Medical History Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Medical History Verbatim Term |
|---|---|---|
| xxxx xxx xxxxx | xxxx xxx xxxx | xxxx |
| | | xxxxxx xxxxxxxxx xx xxxxxx |
| | | xxxxxx xxxxxxxxx xx xxxxx |
| xxxx xxx xxxxx | xxxx xxx xxxxx | xxxx |
| | | xxxxxx xxxxxxxxx xx xxxxxx |
| | | XXXXXX XXXXXXXXX XX XXXXX |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by MedDRA System Organ Class, MedDRA Preferred Term, and Medical History Verbatim Term.

## Listing 16.2.4.2.2: Medical History Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | M: Medical Condition A: Pruritic Condition Associated with Prurigo Nodularis | P: MedDRA Preferred Term<br>S: MedDRA System Organ Class | S: Onset Date<br>E: End Date |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | M: xxxx xxxxxxx (xxxxxxxx xxxxx) A: xxx | P: xxxxxx xxxxxxxxx<br>S: xxxxxxxxxxx | S: xxxx-xx-xx<br>E: |
| | | | M: xxxx xxxxxxx (xxxxxxx xxxxx) A: xxx | P: xxxxxx xxxxxxxxx<br>S: xxxxxxxxxx xxxxxxx | S: xxxx-xx-xx<br>E: |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.

System Organ Class and Preferred Term map to MedDRA (Version 21.1).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Medical Condition/Surgery Verbatim Term, Onset Date, and End Date.

## Listing 16.2.4.3.1: Prurigo Nodularis History Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | Date of Prurigo<br>Nodularis Diagnosis | Body Locations of<br>Prurigo Nodularis | In the 7 days prior to screening, have you had sensation of stinging or burning with your prurigo nodularis? |
|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxx | xxxx-xx-xx | xxxxxxxx xxxxx; xxxxxx; xxxx<br>xxx xxxx; xxxxxxxx | xxx |
| XXXXXX | XXXX | xxxxxxx | xxxx-xx-xx | xxxxxxxx xxxxx; xxxxx xxxxx;<br>xxxxx; xxxxxxxx | xx |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject.

Listing 16.2.4.3.2: Prior Therapies
Treatment Group
(Page xx of yy)

| Subject | Age/Sex | Evaluable | Therapy Type | Name | Estimated<br>Duration (unit) | Route | Reason for<br>Discontinuing Therapy |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxxxxx xxxx | xxxxxxxxxxxx | xx | xxxxxxxxxx | xxxx xx xxxxxxxx |
| | | | xxxxxx xxxxxxx | xxxxx | xxxx | xxxxxxxxxx | xxxxxxxxx |
| | | | xxxx xx xxxxxx<br>xxxxxxx | xxxxxxx xxxxx | xxxxxxxx | xxxxxxxxxxx | xxxxxx |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Therapy Type, Name.

Listing 16.2.4.4.1: Unique Medication Names Coded to WHO DDE ATC Level 2 Terms and Preferred Names (Page xx of yy)

| ATC Level 2 Term | Standardized Medication Name | Medication Name | I: Indication<br>R: Route |
|---|---|---|---|
| ·×××××××××××××××××××××××××××××××××××××× | xxxxxxxxxxx | xxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |
| | | xxxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |
| xxxxxxxxxxx | xxxxxxxxxxx | xxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxxx |
| | | xxxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |

Note: Standardized Medication Name and ATC Level 2 Term map to the WHO DDE (Version September 1, 2018). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by ATC Level 2 Term, Standardized Medication Name, Medication Name, Indication, and Route.

Note to Programmer: If Indication or Route is 'Other' then the applicable variable is 'OTHER: <specification of other>'.

## Listing 16.2.4.4.2: Concomitant Medications Treatment Group (Page xx of yy)

| | | | M: Medication Name | T: Prior/Concomitant | D: Dose |
|---|---|---|---|---|---|
| | | | P: Standardized Medication Name | F: Date of First Dose | U: Units |
| | | | A: ATC Level 2 Term | S: Start Date (Day) 1 | F: Frequency |
| Subject | Age/Sex | Evaluable | I: Indication | E: End Date (Day) 1 | R: Route |
| XXXXXX | XXXX | XXXXXXXXX | M: xxxxxxxxxxx | T: xxxxxxxxx | D: xx |
| | | | P: xxxxxxxxxxxx | F: xxxx-xx-xx | U: xx |
| | | | A: xxxxxxxxxxx | S: xxxx-xx-xx (xx) | F: xxxx |
| | | | I: xxxxxxx | E: xxxx-xx-xx (xx) | R: xxxxxx |
| | | | M: xxxxxxxxxxx | T: xxxxxxxxx | D: xxxxx |
| | | | P: xxxxxxxxxxx | F: xxxx-xx-xx | U: xx |
| | | | A: xxxxxxxxxxx | S: xxxx-xx | F: xx |
| | | | I: xxxxxxx | E: | R: xxxx |
| xxxxxx | xxxx | xxxxxxxxx | M: xxxxxxxxxxx | T: xxxxxxxxx | D: xxx |
| | | | P: xxxxxxxxxxx | F: xxxx-xx-xx | U: xx |
| | | | A: xxxxxxxxxxx | S: xxxx-xx-xx (x) | F: xx |
| | | | I: xxxxxxx | E: xxxx-xx-xx (xx) | R: xxxx |
| | | | ± • * | D. MANA AN AN (AN) | 1/4 1717177 |

Standardized Medication Name and ATC Level 2 Term map to the WHO DDE (Version September 1, 2018).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, Medication Name, Indication, and Route. If ongoing, include 'Ongoing' in place of End Date.

Note to Programmer: If Units, Frequency, Indication, or Route is 'Other' then the applicable variable is 'OTHER: <specification of other>'.

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.

Listing 16.2.4.5: Concomitant Procedures/Therapies
Treatment Group
(Page xx of yy)

| Cubicat | Ago/Sou | Evaluable | T: Procedure/Therapy P: MedDRA Preferred Term | F: Date of First Dose S: Start Date (Day) 1 | Reason for Procedure |
|---|---|---|---|---|---|
| Subject | Age/Sex | Evaluable | S: MedDRA System Organ Class | E: End Date (Day) 1 | or Therapies |
| xxxxxx | xxxx | xxxxxxxxx | T: xxxxxxxxxxxxxxx | F: xxxx-xx-xx | x xxxxxx xxxx xxxxxx |
| | | | P: xxxxxxxxxxxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | xxxxxxxx |
| | | | S: xxxxxxxxxxxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | |
| xxxxx | xxxx | xxxxxxxxx | T: xxxxxxxxxxxxxxx | F: xxxx-xx-xx | x xxxxxx xxxx xxxxxx |
| | | | P: xxxxxxxxxxxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | xxxxxxxx |
| | | | S: xxxxxxxxxxxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | |
| xxxxx | xxxx | xxxxxxxxx | T: xxxxxxxxxxxxxxx | F: xxxx-xx-xx | x xxxxxx xxxx xxxxxx |
| | | | P: xxxxxxxxxxxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | xxxxxxxx |
| | | | S: xxxxxxxxxxxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, and Procedure/Therapy. If ongoing, include 'Ongoing' in place of End Date.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.

System Organ Class and Preferred Term map to MedDRA (Version 21.1).

Listing 16.2.4.6: Physical Examination
Treatment Group
(Page x of xx)

| Subject | Age/Sex | Evaluable | Visit | Date of Assessment (Day) 1 | Physical Exam Completed |
|---|---|---|---|---|---|
| xxxxxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxx-xx-xx (xx) | xxxxxxx |
| xxxxxxxxx | XXXX | xxxxxxxx | xxxxxxxx | xxxx-xx-xx (xx) | xxxxxxxx |
| xxxxxxxxx | xxxx | xxxxxxxx | xxxxxxxx | xxxx-xx-xx (xx) | xxxxxxxx |
| xxxxxxxxx | xxxx | xxxxxxxx | xxxxxxxx | xxxx-xx-xx (x) | xxxxxxxx |
| xxxxxxxxx | xxxx | xxxxxxxx | xxxxxxxx | xxxx-xx-xx (xx) | xxxxxxx |
| XXXXXXXXX | XXXX | XXXXXXXX | XXXXXXXXX | xxxx-xx-xx (xx) | XXXXXXX |

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
 date - date of first dose + 1 for dates on or after first dose.
Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.5.1: Study Visit/Phone Call Compliance
Treatment Group
(Page xx of yy)

| Subject | Age/Sex | Evaluable | · Visit | Visit Date | Study<br>Day¹ | Visit | Continuing into MTI-107? | Visit Not Done/<br>Reason for Unscheduled Visit |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxx-xx-xx | xx | xxx | xxx | |
| | | | xxxxxxx | xxxx-xx-xx | xx | xxx | xxx | |
| | | | xxxxxx | xxxx-xx-xx | xx | xxx | xxx | |
| | | | xxxxxx | xxxx-xx-xx | XX | XXX | xxx | xxxxxxx x xxxxxx xxxxxx xxxxx xxxxx xxxx |
| | | | xxxxxx | xxxx-xx-xx | xx | xxx | xxx | |
| | | | xxxxxxxxxxxx | xxxx-xx-xx | XX | XXX | xxx | |
| xxxxxx | XXXX | xxxxxxx | xxxxxxxx | xxxx-xx-xx | XX | xxx | xxx | |
| | | | xxxxxx | xxxx-xx-xx | xx | xxx | xxx | |
| | | | xxxxxxxxxxxx | xxxx-xx-xx | XX | xxx | xxx | |

Listing sorted by Subject, Visit, and Visit Date.

Note to Programmer: If a visit is ranged present the 'Visit Date' column as '<Start Date> to <End Date>' same with the Study Day column.

<sup>1</sup> Day is calculated as date - baseline date for dates prior to baseline date. Otherwise, day is calculated as
 date - baseline date + 1 for dates on or after baseline date. For follow-up visits, Week 10 date is used in place of baseline.
Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.5.2: Study Drug Dispensing and Return
Treatment Group
(Page xx of yy)

| Subject | Age/Sex | Evaluable | Bottle<br>Number | Date Bottle<br>Dispensed | Date Bottle<br>Returned | Number of Tablets<br>Dispensed | Number of Tablets<br>Returned | Tablets Used |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxx | xxxx-xx-xx<br>xxxx-xx-xx | xxxx-xx-xx | xx<br>xx | xx<br>xx | xx<br>xx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxx | xxxx-xx-xx<br>xxxx-xx-xx | xxxx-xx-xx | xx<br>xx | xx<br>xx | xx<br>xx |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Date Bottle Dispensed, and Date Bottle Returned.

## Listing 16.2.5.3: Dosing Deviations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | Date of Deviation | Reason for Deviation | Number of Tablets Taken |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxx-xx-xx | xxxxxx | xxxxxxxxxxxxxxxxx |
| xxxxx | xxxx | xxxxxxxx | xxxx-xx-xx<br>xxxx-xx-xx | xxxxxx | x<br>xxxxxxxxxxxxxxxxxx |
| | | | xxxx-xx-xx | xxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| xxxxxx | XXXX | XXXXXXXX | xxxx-xx-xx<br>xxxx-xx-xx | xxxx<br>xxxxxx | x |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Date of Deviation, Type of Deviation, and Number of Tablets Taken.

Listing 16.2.6.1.1: Worst Itch Numeric Rating Scale (WI-NRS) at Screening Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | Date of Assessment (Day) <sup>1</sup> | WI-NRS <sup>2</sup> in the past 24 hours |
|---|---|---|---|---|
| xxxxxxx | xxxx | xxxxxxxx | xxxx-xx-xx (xx) | XX |
| xxxxxxx | xxxx | xxxxxxxx | xxxx-xx-xx (xx) | xx |
| xxxxxxx | xxxx | xxxxxxxx | xxxx-xx-xx (xx) | xx |
| xxxxxxx | xxxx | xxxxxxxx | xxxx-xx-xx (xx) | XX |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>&</sup>lt;sup>2</sup> Scaled from 0 - No Itch to 10 - Worst Itch Imaginable.

Listing 16.2.6.1.2: Worst Itch Numeric Rating Scale (WI-NRS)

Treatment Group

(Page xx of yy)

| Subject | Age/Sex | Evaluable | Timepoint | Date of Assessment ( | Day) ¹ | WI-NRS in past 24 hrs² | Change from<br>Baseline <sup>3</sup> |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | | xxxx-xx-xxTxx:xx | (xxx) | х | |
| | | | | xxxx-xx-xxTxx:xx:xx | (xxx) | X | |
| | | | | xxxx-xx-xxTxx:xx:xx | (xxx) | X | |
| | | | | xxxx-xx-xxTxx:xx:xx | (xxx) | X | |
| | | | | xxxx-xx-xxTxx:xx:xx | (xxx) | X | |
| | | | | xxxx-xx-xxTxx:xx:xx | (xxx) | X | |
| | | | xxxxxxx | xxxx-xx-xxTxx:xx:xx | (xxx) | X | |
| | | | XXXXXXX | xxxx-xx-xxTxx:xx | (XXX) | X | |
| | | | XXXXXXX | xxxx-xx-xxTxx:xx | (XXX) | X | |
| | | | XXXXXXX | xxxx-xx-xxTxx:xx | (XXX) | X | |
| | | | XXXXXXX | Average | (11111) | XXXXX | |
| | | | | - | | | |
| | | | xxxxxxx | xxxx-xx-xxTxx:xx:xx | (xxx) | X | XXXX |
| | | | XXXXXXX | xxxx-xx-xxTxx:xx:xx | (xxx) | X | XXXX |
| | | | XXXXXXX | xxxx-xx-xxTxx:xx:xx | (xxx) | X | XXXX |
| | | | XXXXXXX | xxxx-xx-xxTxx:xx:xx | (xxx) | X | XXXX |
| | | | XXXXXXX | Average | | XXXXX | XXXX |

Listing sorted by Subject, Date of Assessment, Timepoint (where the Average over a given Timepoint is presented in the order above), and WI-NRS in past 24 hours.

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>&</sup>lt;sup>2</sup> Scaled from 0 - No Itch to 10 - Worst Itch Imaginable

<sup>&</sup>lt;sup>3</sup> The WI-NRS Baseline is the average of the results for the week prior to starting the study drug (Timepoint = BASELINE). Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.6.2: IGA PN-A and IGA PN-S Results
Treatment Group
(Page xx of yy)

| Subject | Age/Sex | Evaluable | Visit | Date of Assessment (Day) 1 | Investigator's Global Assessement of Prurigo Nodularis Activity | Investigator's Global Assessement of Prurigo Nodularis Stage |
|---|---|---|---|---|---|---|
| xxxxxxx | xxxx | xxxxxxxx | xxxxxxx | xxxx-xx-xx (xx) | XXXXX X | xxxxx x |
| | | | | xxxx-xx-xx (xx) | xxxxx x | xxxxx x |
| | | | | xxxx-xx-xx (xx) | xxxxx x | xxxxx x |
| | | | | xxxx-xx-xx (xx) | xxxxx x | xxxxx x |
| | | | | xxxx-xx-xx (xx) | xxxxx x | xxxxx x |
| | | | | xxxx-xx-xx (xx) | xxxxx x | xxxxx x |
| xxxxxxx | xxxx | xxxxxxxx | xxxxxx | xxxx-xx-xx (xx) | xxxxx x | xxxxx x |
| | | | | xxxx-xx-xx (xx) | xxxxx x | xxxxx x |
| | | | | xxxx-xx-xx (xx) | xxxxx x | xxxxx x |
| | | | | xxxx-xx-xx (xx) | xxxxx x | XXXXX X |
| | | | | xxxx-xx-xx (xx) | XXXXX X | XXXXX X |
| | | | | xxxx-xx-xx (xx) | XXXXX X | XXXXX X |

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
 date - date of first dose + 1 for dates on or after first dose.
Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

## Listing 16.2.6.3: Dermatology Life Quality Index (DLQI) Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | Visit<br>Date of Assessment | (Day) 1 | Question<br>Number | | Result |
|---|---|---|---|---|---|---|---|
| xxxxxxx xxxx | xxxxxx | xxxxxxxxx<br>xxxx-xx-xx (xx) | | 1 | Over the last week, how itchy, sore, painful or stinging has your skin been? | xxxxx | |
| | | | | | 2 | Over the last week, how embarrassed or self conscious have you been because of your skin? | xxxxxx |
| | | | | 3 | Over the last week, how much has your skin interfered with you going shopping or looking after your home or garden? | xxxxxx | |
| | | | | 4 | Over the last week, how much has your skin influenced the clothes you wear? | XXXXXX | |
| | | | | 5 | Over the last week, how much has your skin affected any social or leisure activities? | XXXXXX | |
| | | | | | 6 | Over the last week, how much has your skin made it difficult for you to do any sport? | xxxxxx |
| | | | | | 7 | Over the last week, has your skin prevented you from working or studying? | XXXXXX |
| | | | | | 7A | If "No", over the last week how much has your skin been a problem at work or studying? | xxxxxx |
| | | | | | 8 | Over the last week, how much has your skin created problems with your partner or any of your close friends or relatives? | xxxxx |
| | | | | 9 | Over the last week, how much has your skin caused any sexual difficulties? | XXXXXX | |
| | | | | | 10 | Over the last week, how much of a problem has the treatment for your skin been, for example by making your home messy, or by taking up time? | xxxxxx |
| | | | | | | Questionnaire Score | XX |

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.6.4: Photography
Treatment Group
(Page xx of yy)

| Subject | Age/Sex | | Visit<br>Date of Ass | sessment (Day)¹ | Body Area: | s Photographed | d |
|---|---|---|---|---|---|---|---|
| xxxxxxx | XXXX | xxxxxx | xxxxxxxxx<br>xxx-xx-xx | (xx) | xxxxxxxx; | xxxxxxxxx; | xxxxxxxx |
| | | | xxxxxxxxx<br>xxx-xx-xx | (xx) | xxxxxxxx; | xxxxxxxxx; | xxxxxxxx |
| | | | xxxxxxxxx<br>xxx-xx-xx | (xx) | xxxxxxx; | xxxxxxxxx; | xxxxxxx |
| | | | xxxxxxxx<br>xxx-xx-xx | | xxxxxxx; | xxxxxxxxxx; | xxxxxxxx |

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
 date - date of first dose + 1 for dates on or after first dose.
Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.7.1.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| ************************************** | | | |
|---|---|---|---|
| ************************************** | MedDRA System Organ Class | MedDRA Preferred Term | Adverse Event |
| ************************************** | xxxxx xxxxx xxxxx | XXXXX XXXXX XXXXX | xxxxxxxxx |
| ************************************** | | | xxxxxxx xxxxxxx xxxxxxxx |
| ************************************** | | | xxxxxxxx xxxxxxxx xxxxxxxxxxxxxxx |
| ************************************** | | xxxxx xxxxx xxxxx | xxxxxxxxx |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | xxxxxxx xxxxxxx xxxxxxxx |
| xxxxxxxx xxxxxxxx xxxxxxxxxxxxxxxxxxxx | | | xxxxxxxx xxxxxxxx xxxxxxxxxxxxxxx |
| | | xxxxxxxxx | xxxxx xxxxx xxxxx |
| ******** ******** ******************** | | | xxxxxxx xxxxxxx xxxxxxxx |
| AAAAAAAAA AAAAAAAAA | | | ******** ******* ********* |

Note: System Organ Class and Preferred Term map to MedDRA (Version 21.1).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by MedDRA System Organ Class, Preferred Term, and Adverse Event.

## Listing 16.2.7.1.2: Treatment-Emergent Adverse Events Treatment Group (Page xx of yy)

| | | | | S: Is AE Serious? |
|---|---|---|---|---|
| | | | S: Grade <sup>2</sup> | R: Reason(s) for Serious |
| S: Subject | A: Event | F: Date of First Dose | R: Relationship to Study | T: Action Taken with |
| A: Age/Sex | C: System Organ Class | S: Start Date (Day) 1 | Treatment | Study Treatment |
| E: Evaluable | P: Preferred Term | E: End Date (Day) 1 | O: Outcome | A: Any Other Action(s) |
| S: xxxxxx | A: xxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxx xxx xxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |
| | A: xxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (x) | R: xxxxxxxxxx | R: xxxx xxx xxxxxx |
| | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |
| S: xxxxxx | A: xxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxx xxx xxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |
| S: xxxxxx | A: xxxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxx xxx xxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |

System Organ Class and Preferred Term map to MedDRA (Version 21 SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, and Adverse Event.

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>2</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.
Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
System Organ Class and Preferred Term map to MedDRA (Version 21.1).

## Listing 16.2.7.1.3: Serious Adverse Events Treatment Group (Page xx of yy)

| | | | | S: Is AE Serious? |
|---|---|---|---|---|
| | | | S: Grade <sup>2</sup> | R: Reason(s) for Serious |
| S: Subject | A: Event | F: Date of First Dose | R: Relationship to Study | T: Action Taken with |
| A: Age/Sex | C: System Organ Class | S: Start Date (Day) 1 | Treatment | Study Treatment |
| E: Evaluable | P: Preferred Term | E: End Date (Day) <sup>1</sup> | O: Outcome | A: Any Other Action(s) |
| S: xxxxxx | A: xxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxx xxx xxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |
| | A: xxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (x) | R: xxxxxxxxxx | R: xxxx xxx xxxxxx |
| | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |
| S: xxxxxx | A: xxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxx xxx xxxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |
| S: xxxxxx | A: xxxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxx xxx xxxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.

System Organ Class and Preferred Term map to MedDRA (Version 21.1).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, and Adverse Event.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>&</sup>lt;sup>2</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.

Listing 16.2.7.1.4: Subjects Who Permanently Discontinued Study Drug Due to Adverse Events

Treatment Group

(Page xx of yy)

| | | Completion/Discontinuation | | lverse Events |
|---|---|---|---|---|
| | F: Date of First | T: Primary Reason for Treatment | A: Event | S: Start Date (Day) 1 |
| S: Subject | Dose | Discontinuation | S: Grade <sup>2</sup> | E: End Date (Day) 1 |
| A: Age/Sex | L: Date of Last | S: Primary Reason for Study | R: Relationship to | A: Action Taken with Study |
| E: Evaluable | Dose | Discontinuation | Study Treatment | Treatment |
| S: xxxxx | F: xxxx-xx-xx | D: xxxx-xx-xx (xx) | A: xxxxxxxxx | S: xxxx-xx-xx (xx) |
| A: xxxx | L: xxxx-xx-xx | T: xxxxxx | S: xxxxxxx | E: xxxx-xx-xx (xx) |
| E: xxxxxxx | | S: xxxxxxxxxxxx | R: xxxxxxxxxxxxxxx | A: xxxxxxxxxxx |

Listing sorted by Subject, Start Date, End Date, and Adverse Event.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>2</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.
Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.7.2.1: Hospital Anxiety and Depression Scale

Treatment Group

(Page xx of yy)

V: Visit
Subject Age/Sex Evaluable D: Date of Assessment (Day) Question Result

XXXXXXXX XXXX xxxxxxx V: xxxxxxxxx I feel tense or 'wound up' xxxxxxxxxxxxxxxx I still enjoy the things I used to enjoy D: xxxx-xx-xx (xx) xxxxxxxxxxxxxxxx I get a sort of frightened feeling as if something awful is about to happen xxxxxxxxxxxxxxxxx I can laugh and see the funny side of things xxxxxxxxxxxxxx Worrying thoughts go through my mind XXXXXXXXXXXXXXXXXX I feel cheerful XXXXXXXXXXXXXXXXXX I can sit at ease and feel relaxed xxxxxxxxxxxxxxxx Depression Subscale Anxiety Subscale

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.7.2.2: Epworth Sleepiness Scale
Treatment Group
(Page xx of yy)

V: Visit Subject Age/Sex Evaluable D: Date of Assessment (Day) 1 Situation Result XXXXXXXX XXXX xxxxxxx V: xxxxxxxxx Sitting and reading xxxxxxxxxxxxxxxxx Watching TV D: xxxx-xx-xx (xx) XXXXXXXXXXXXXXXXXX Sitting, inactive in a public place (e.g. a theatre or a meeting) XXXXXXXXXXXXXXXXX As a passenger in a car for an hour without a break xxxxxxxxxxxxxxxxx Lying down to rest in the afternoon when circumstances XXXXXXXXXXXXXXXXXX Sitting and talking to someone xxxxxxxxxxxxxxxxx Sitting quietly after a lunch without alcohol XXXXXXXXXXXXXXXXXX In a car, while stopped for a few minutes in the

traffic

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

XXXXXXXXXXXXXXXXXX

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.

Listing 16.2.7.3: Menstrual Diary
Treatment Group
(Page xx of yy)

| Subject Age/Sex Evaluable | Childbearing Potential | Start Date of Period (Day)¹ | End Date of Period (Day) 1 |
|---|---|---|---|
| xxxxxxx xxxx xxxxx | xxxxxxxxxxx | xxxx-xx-xx (xx)<br>xxxx-xx-xx (xx)<br>xxxx-xx-xx (xx) | xxxx-xx-xx (xx)<br>xxxx-xx-xx (xx) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.

## Listing 16.2.8.1: Pregnancy Test Results Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Evaluable | V: Visit<br>D: Date (Day) <sup>1</sup> | S: Specimen <sup>2</sup><br>R: Result | S: Was a Serum Pregnancy Test Ordered? E: If no, but was required, explain | Comments |
|---|---|---|---|---|
| S: xxxxx | V: xxxxxxxx | S: xxxx | S: xxx | ********** |
| A: xxxx<br>E: xxxxxxxx | D: xxxx-xx-xx (xxx) | R: xxxxxxxx | E: | ΑΛΛΑΛΑΛΑΛΑΛΑΛΑ |
| | V: xxxxxxxx | S: xxxxx | S: xx | |
| | D: xxxx-xx-xx (xxx) | R: xxxxxxxx | E: | |
| | V: xxxxxxxx | S: xxxxx | S: xx | |
| | D: xxxx-xx-xx (xxx) | R: xxxxxxxx | E: | |
| | V: xxxxxxxx | S: xxxxx | S: xx | |
| | D: xxxx-xx-xx (xxx) | R: xxxxxxxx | E: | |
| S: xxxxxx | V: xxxxxxxx | S: xxxxx | S: xx | |
| A: xxxx<br>E: xxxxxxx | D: xxxx-xx-xx (xxx) | R: xxxxxxxx | E: xxxxxxxxxxxxxxxxxxxxxxx | |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date, and Specimen. NOTE: Serum Pregnancy Questions (S: E:) are only applicable to Urine Pregnancy test records.

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>&</sup>lt;sup>2</sup> For Serum pregnancy results: HCG levels less than 10 mIU/mL are considered negative for pregnancy. Levels between 10 - 24.9 mIU/mL are equivocal and a redraw of the patient after 48 hours is suggested. Levels greater than or equal to 25 mUI/mL are considered positive for pregnancy.

## Listing 16.2.8.2.1: Laboratory Test Results Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex | V: Visi | | | Results | | | Refe | rence Range | | |
|---|---|---|---|---|---|---|---|---|---|---|
| E: Evaluable | C: Cate | egory | Laboratory Test | (Units) | Ī | Low | High | Indicator (CS | 52) | Comments |
| | V: xxxx | | ****** | xxxx (xx | (xxxx) | | | | | ***** |
| : xxxxxxxx | | x-xx-xxTxx:xx:xx (xxx)<br>xxxxxxxxxxxxxxxx | | | | | | | | xxxxxxxxxxxxxxxxxx |
| | | xxxxxx<br>x-xx-xxTxx:xx:xx (xxx)<br>xxxxxxxxxxxxxxxx | ********* | xxxx (xx | xxxx) | X | xx | xxxxxxxxx | (xxx) | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | xxxxx<br>x-xx-xxTxx:xx:xx (xxx)<br>xxxxxxxxxxxxxx | ××××××××××××××××××××××××××××××××××××××× | xxxx (xx | xxxx) x | K | xx | xxxxxxxxx | (xxx) | |

Listing sorted by Subject, Visit, Date, Category, and Lab Test.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>&</sup>lt;sup>2</sup> Clinical significance based on Investigator interpretation. CS = Clinically Significant; NCS = Not Clinically Significant. Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.8.2.2: Out of Range Laboratory Results
Treatment Group
(Page xx of yy)

| A: Age/Sex | V: Visit D: Date (Day) 1 | | Results | | | rence Range | - |
|---|---|---|---|---|---|---|---|
| E: Evaluable | C: Category | Laboratory Test | (Units) | Low | High | Indicator (CS2) | Comments |
| S: xxxxx<br>A: xxxx<br>E: xxxxxxx | V: xxxxxxxxx D: xxxx-xx-xxTxx:xx:xx (xxx) C: xxxxxxxxxxxxxxxxxxxx | ******** | xxxx (xxxxxx) | | | | ************************************** |
| | V: xxxxxxxxx D: xxxx-xx-xxTxx:xx:xx (xxx) C: xxxxxxxxxxxxxxxxxxxxx | *********** | xxxx (xxxxxx) | х | xx | xxxxxxxxxx (xxx) | ************************************** |
| | V: xxxxxxxx<br>D: xxxx-xx-xxTxx:xx:xx (xxx)<br>C: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | ********* | xxxx (xxxxxx) | Х | xx | xxxxxxxxxx (xxx) | |

Listing sorted by Subject, Visit, Date, Category, and Lab Test.

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>&</sup>lt;sup>2</sup> Clinical significance based on Investigator interpretation. CS = Clinically Significant; NCS = Not Clinically Significant. Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.8.2.3: Common Laboratory Comments Including Reference Ranges for Specific Laboratory Tests (Page 1 of 1)

| <del></del> | | |
|---|---|---|
| Category | Laboratory Test | Comments |
| xxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxx | *************************************** |
| | | *************************************** |
| | xxxxxxxxxxxxxxxxxx | *************************************** |
| | | ***************************** |
| | | *************************************** |
| | | ************************* |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| xxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxx | *************************************** |
| | | ************************** |
| | | ***************************** |
| | | ******************* |
| | | *************************************** |
| xxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxx | *************************************** |
| | | ***************************** |
| | | *************************************** |
| | | *************************************** |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Category and Lab Test.

Listing 16.2.8.3: Electrocardiogram Test Results

Treatment Group

(Page x of xx)

| S: Subject<br>A: Age/Sex<br>E: Evaluable | Category ECG Parameter | V: Visit<br>D: Date/Time of ECG (Day) <sup>1</sup> | Result (unit) | Clinical<br>Significance <sup>2</sup> | Comments |
|---|---|---|---|---|---|
| S: xxxxxxxx<br>A: xxxx | xxxxxxxxx xxxxxxxx | V: xxxxxxxx<br>D: xxxx-xx-xxTxx:xx (xx) | xxxx xxxxx xx (xxx) | xxx | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

E: xxx/xx/xxx

Listing sorted by Subject, Category, Parameter, Visit, and Date. Note: for interpretation records, EGEVAL should be concatenated into ECG Parameter as EGTEST (EGEVAL).

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as

date - date of first dose + 1 for dates on or after first dose.

<sup>2</sup> Clinical significance based on Investigator interpretation. CS = Clinically Significant; NCS = Not Clinically Significant.

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.

Listing 16.2.8.4: Vital Signs
Treatment Group
(Page x of xx)

| Subject | Age/Sex | Evaluable | Visit | Date of Measurements (Day) 1 | Vital Sign | Result | Units |
|---|---|---|---|---|---|---|---|
| xxxxxxx | VVVV | xxxxx | xxxxxxxxx | xxxx-xx-xx (xxx) | xxxxx xxx | XX | xxxx |
| | ΔΛΛΛ | ΑΛΛΛΛ | ΑΛΛΑΛΑΛΑΛ | AAAA AA AA (AAA) | XXXXX XXX | XX | XXXX |
| | | | | | XXXXX XXX | XX | XXXX |
| | | | | | XXXXX XXX | XX | XXXX |
| | | | | | XXXXX XXX | XX | XXXX |
| | | | xxxxxxxxx | xxxx-xx-xx (xxx) | XXXXX XXX | XX | xxxx |
| | | | | | xxxxx xxx | xx | XXXX |
| | | | | | xxxxx xxx | xx | XXXX |
| | | | | | xxxxx xxx | xx | XXXX |
| | | | | | XXXXX XXX | XX | XXXX |
| xxxxxxx | xxxx | xxxxx | xxxxxxxxx | xxxx-xx-xx (xxx) | XXXXX XXX | XX | xxxx |
| | | | | , , | xxxxx xxx | XX | xxxx |
| | | | | | xxxxx xxx | XX | xxxx |
| | | | | | xxxxx xxx | XX | xxxx |
| | | | | | xxxxx xxx | xx | xxxx |
| | | | xxxxxxxxx | xxxx-xx-xx (xxx) | XXXXX XXX | XX | xxxx |
| | | | | ,, | XXXXX XXX | XX | XXXX |
| | | | | | XXXXX XXX | XX | XXXX |
| | | | | | XXXXX XXX | XX | XXXX |
| | | | | | XXXXX XXX | XX | XXXX |

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date, and Vital Sign (ordered as: Height, Weight, Temperature, Respiration Rate, Heart Rate, Systolic Blood Pressure, Diastolic Blood Pressure).

Listing 16.2.8.5: Pharmacokinetics Blood Sample Collection and Plasma Concentrations Treatment Group  $(Page \ x \ of \ xx)$ 

| S: Subject<br>A: Age/Sex<br>A: Evaluable | Analyte | Visit | Date/Time of Pre-PK<br>Study Drug Dose | Date/Time PK<br>Sample Obtained | Concentration (ng/mL) | Reason Not Done |
|---|---|---|---|---|---|---|
| 3: xxxxx<br>A: xxxx | xxxxxxxxx | xxxxxxxxx | xxxx-xx-xxTxx:xx | xxxx-xx-xxTxx:xx | xxxxxxxxx | xxxxxxxx |
| | | xxxxxxxxx | xxxx-xx-xxTxx;xx | xxxx-xx-xxTxx;xx | xxxxxxxxx | xxxxxxxx |
| | | xxxxxxxxx | xxxx-xx-xxTxx:xx | xxxx-xx-xxTxx:xx | xxxxxxxxx | xxxxxxxx |
| | | xxxxxxxxx | xxxx-xx-xxTxx:xx | xxx-xx-xxTxx;xx | xxxxxxxxx | xxxxxxxx |
| | xxxxxxxxx | xxxxxxxxx | xxxx-xx-xxTxx:xx | xxxx-xx-xxTxx:xx | xxxxxxxxx | xxxxxxxx |
| | | xxxxxxxxx | xxxx-xx-xxTxx:xx | xxxx-xx-xxTxx:xx | xxxxxxxxx | xxxxxxxx |
| : xxxxx<br>: xxxx | xxxxxxxxxx | xxxxxxxxx | xxxx-xx-xxTxx;xx | xxxx-xx-xxTxx:xx | xxxxxxxxx | xxxxxxxx |
| | | xxxxxxxxx | xxxx-xx-xxTxx:xx | xxxx-xx-xxTxx:xx | xxxxxxxxx | xxxxxxxx |
| | | xxxxxxxxx | xxxx-xx-xxTxx;xx | xxxx-xx-xxTxx;xx | xxxxxxxxx | xxxxxxxx |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Analyte, Visit, Date.